

Protocol No.: APL2-202

A Phase IIa, Open Label, Multiple Dose Study to Assess the Safety, Efficacy and Pharmacokinetics of Subcutaneously Administered APL-2 in Subjects with Paroxysmal Nocturnal Hemoglobinuria (PNH)

Phase: Ila

Version: Protocol Version 3.0

Date: 31 January 2018

EudraCT No: 2017-005140-16

## **Confidentiality Statement**

This document is confidential. It contains proprietary information of Apellis Pharmaceutical, Inc. Any viewing or disclosure of such information that is not authorized in writing by Apellis Pharmaceutical, Inc is strictly prohibited. Such information may be used solely for the purpose of reviewing or performing this study.

# **SIGNATURE PAGE**

Protocol APL2-202 was approved by:



Apellis Pharmaceuticals

| A Phase IIa, Open Label, Multiple Dose Study to Assess the Safety, Efficacy and Pharmacokinetics of Subcutaneously Administered APL-2 in Subjects with Paroxysmal Nocturnal Hemoglobinuria (PNH) Protocol Number, Version and Date: Study Phase: Study Phase: Phase IIa Apellis Pharmaceuticals 6400 Westwind Way, Suite A Crestwood, KY 40014 Investigational Test Article: Indication Studied: PNH Investigator Agreement: I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practices (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, and all applicable regulatory requirements. Principal Investigator: Name: Signature: Date: Date: (DD/MMM/YYYY) | INVESTIGATOR AGREEMENT | |
|---|---|---|
| Study Phase: Sponsor Name and Address: Apellis Pharmaceuticals 6400 Westwind Way, Suite A Crestwood, KY 40014 Investigational Test Article: Indication Studied: PNH Investigator Agreement: I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practices (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, and all applicable regulatory requirements. Principal Investigator: Name: Signature: | Long Title: | Assess the Safety, Efficacy and Pharmacokinetics of Subcutaneously Administered APL-2 in Subjects |
| Sponsor Name and Address: Apellis Pharmaceuticals 6400 Westwind Way, Suite A Crestwood, KY 40014 Investigational Test Article: APL-2 Indication Studied: PNH Investigator Agreement: I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practices (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, and all applicable regulatory requirements. Principal Investigator: Name: Signature: Signature: | | APL2-202/Version 3.0/31Jan2018 |
| 6400 Westwind Way, Suite A Crestwood, KY 40014 Investigational Test Article: Indication Studied: Investigator Agreement: I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practices (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, and all applicable regulatory requirements. Principal Investigator: Name: Signature: | Study Phase: | Phase IIa |
| Investigator Agreement: I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practices (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, and all applicable regulatory requirements. Principal Investigator: Name: Signature: | Sponsor Name and Address: | 6400 Westwind Way, Suite A |
| I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practices (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, and all applicable regulatory requirements. Principal Investigator: Name: Signature: | Investigational Test Article: | APL-2 |
| recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practices (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, and all applicable regulatory requirements. Principal Investigator: Name: Signature: | Indication Studied: | PNH |
| Signature: | Investigator Agreement: | recognize its confidentiality, and agree to conduct<br>the described trial in compliance with Good Clinical<br>Practices (GCP), the ethical principles contained<br>within the Declaration of Helsinki, this protocol, and |
| | Principal Investigator: | Name: |
| Date:/(DD/MMM/YYYY) | | Signature: |
| | | Date:/(DD/MMM/YYYY) |

# **TABLE OF CONTENTS**

| | ABLE OF CONTENTS | |
|-----|--------------------------------------------------------|----|
| LIS | ST OF TABLES | 7 |
| 1. | SYNOPSIS | 8 |
| 2. | STUDY FLOW CHART | 13 |
| 3. | ABBREVIATIONS | |
| 4. | INTRODUCTION | 20 |
| | 4.1 Background | |
| | 4.1.1 Paroxysmal Nocturnal Hemoglobinuria | |
| | 4.1.2 APL-2 | |
| | 4.1.3 Nonclinical Data | |
| | 4.1.3.1 Pharmacology | |
| | 4.1.3.2 Pharmacokinetics | |
| | 4.1.3.3 Toxicology | |
| | 4.1.4 Clinical Data | |
| | 4.1.6 Ongoing Clinical Studies III Healthy Volunteers | |
| | 4.2 Rationale | |
| | 4.2.1 Purpose of the Study | |
| | 4.2.2 Dose Selection | |
| | 4.3 Risk/Benefit | |
| 5. | | |
| J. | 5.1 Study Objectives | |
| | 5.2 Study Endpoints | |
| 6. | | |
| 7. | | |
| • | 7.1 Inclusion Criteria | |
| | 7.1.1 Approved methods of contraception | |
| | 7.2 Exclusion Criteria | |
| 8. | STUDY TREATMENTS | |
| | 8.1 Allocation to Treatment | |
| | 8.2 Blinding | |
| | 8.3 Treatments Administered | |
| | 8.3.1 Drug supplies | 31 |
| | 8.3.1.1 Identity of Investigational Products | |
| | 8.3.1.2 Study Supplies | 31 |
| | 8.3.1.3 Accountability | |
| | 8.3.2 Planned Dose Levels and Dosing Schedule | |
| | 8.3.3 Drug Administration | |
| | 8.4 Concomitant Medications | |
| | 8.4.1 Prophylactic antibiotics | |
| | 8.4.1.1 Primary prophylactic antibiotic Day 1-14 | |
| | 8.4.1.2 Primary prophylactic antibiotic Day 15 onwards | |
| | 8.4.1.3 Alternative prophylactic antibiotics | |
| | 8.4.2 Rescue antibiotics 8.4.3 Vaccinations | |
| | 8.4.4 Iron Supplements | |
| | 8.4.5 Phlebotomy/Venesection for iron overload | |
| 9. | · | |
| ٥. | 9.1 Screening | |
| | 0.1 0.100/m/g | |

| | 9.2 | Part 1 | 1 - Treatn | nent Period – (Days 1 to 28) | 34 |
|---|---|---|---|---|---|
| | | 9.2.1 | On Site | Administration (Day 1 to Day 3 and Days 8, 15 and 22) | 34 |
| | | 9.2.2 | Outpatie | ent Administration (Day 4 to Day 28) | 34 |
| | 9.3 | Part 2 | 2A - Trea | tment Period – (Days 29 to 84) | 34 |
| | | 9.3.1 | On Site | Administration (Days 29, 36, 43, 57 and 71) | 34 |
| | | 9.3.2 | | ent Administration (Day 30 to Day 84) | |
| | 9.4 | Part 2 | 2B - Trea | tment Period – (Days 85 to 364) | 35 |
| | | 9.4.1 | | Administration (Days 85, 113, 141, 169, 197, 225, 253, 281, 309, ar | |
| | | 9.4.2 | • | ent Administration (Day 85 to Day 364) | |
| | | | | /-up - (Days 365, 379, and 393) | |
| | | 9.5.1 | | it (Day 414, or Day 134, or Day 78) | |
| | | 9.5.2 | | duled Follow-up Visits | |
| | | 9.5.3 | | led End of Study | |
| | | | | y Review | |
| | | 9.6.1 | • | Monitoring Committee | |
| 40 | 9.7 | | | ubjects from the Study | |
| 10. | | | | | |
| | | | | ************************************** | |
| | | | • | eight and Weight | |
| | | | • | I Examination | |
| | | | | jns | |
| | | | | cardiogram Monitoringnal Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale | |
| | | | | Analog Scale Assessment (LASA) for Quality of Life | |
| | | | | Laboratory Tests | |
| | | | ).1.7.1 | Hematology | |
| | | | ).1.7.2 | Coagulation | |
| | | | 0.1.7.3 | Serum Chemistry | |
| | | | ).1.7.4 | Urinalysis | |
| | | 10 | .1.7.5 | Human Chorionic Gonadotropin (Serum Pregnancy Test) and Foll | |
| | | | | Stimulating Hormone | 39 |
| | | 10.1.8 | Injection | n/ Infusion Site and Pump Safety Assessment | 39 |
| | | | | tic Assessments | |
| | | | | ampling and Processing | |
| | | | | al Method | |
| | | | • | ry Assessments | |
| | | | | amic Assessments | |
| | | | | ntibody Assessment | |
| | | | | for Study Assessments | |
| | | _ | - | ts | |
| 11. | | | | S | |
| | | | | verse Events | |
| | | | | f Adverse Events | |
| | | | | / | |
| | | | | ty | |
| | | | | Adverse Event | |
| | | | | ious Adverse Event | |
| | | | | ts of Special Interest | |
| | 11.6 | Unex | pected A | dverse Events or Unexpected Suspected Adverse Reactions | 45 |

| | 11.7 Treatment and Follow up of Adverse Events | 45 |
|---|---|---|
| | 11.8 Pregnancy | |
| 12 | STATISTICS | |
| 12. | 12.1 Sample Size Justification | |
| | 12.2 Statistical Analysis Methodology | |
| | 12.2.1 Analysis Populations | |
| | 12.2.1.1 Screened Population | |
| | 12.2.1.3 Pharmacokinetic (PK) Population | |
| | 12.2.1.5 Data Review for Analysis Populations | |
| | 12.2.2 Study Endpoints | |
| | 12.2.2.1 Safety Endpoints | |
| | 12.2.2.2 Efficacy Endpoints | |
| | 12.2.2.3 Secondary Endpoints | |
| | 12.2.2.4 Pharmacokinetic Endpoints | |
| | 12.2.2.5 Exploratory Pharmacodynamic Endpoints (Markers) | |
| | 12.2.3 Safety Analyses | |
| | 12.2.3.1 Adverse Events | |
| | 12.2.3.2 Clinical Laboratory Tests | |
| | 12.2.3.3 Vital Signs and ECGs | |
| | 12.2.4 Efficacy and Secondary Endpoint Analyses | |
| | 12.2.5 Pharmacokinetic Analyses | |
| | 12.2.6 Pharmacodynamic Analyses | |
| | 12.2.7 Handling of Dropouts and/or Missing Data | |
| | 12.2.8 Other Data Analyses | |
| | · | |
| 40 | 12.3 Interim Analyses | |
| 13. | ADMINISTRATIVE CONSIDERATIONS | |
| | 13.1 Direct Access to Source Data/Documents | |
| | 13.2 Quality Control and Quality Assurance | |
| | 13.2.1 Monitoring | |
| | 13.3 Ethics | |
| | 13.3.1 Ethical Conduct of the Study | |
| | 13.3.2 Institutional Review Board/Ethic Committee | |
| | 13.3.3 Subject Information and Consent | |
| | 13.3.4 Confidentiality | |
| | 13.3.5 ClinicalTrials.gov | |
| | 13.3.6 Termination of Study | |
| | 13.4 Data Handling and Record Keeping | 50 |
| | 13.5 Protocol Amendments | 51 |
| | 13.6 Report Format | 51 |
| | 13.7 Finance and Insurance | |
| | 13.8 Publication Policy | |
| 14. | REFERENCES | |
| | APPENDIX 1: FUNCTIONAL ASSESSMENT OF CHRONIC ILLNESS THERAPY (FACIT) | |
| | FATIGUE SCALE | 53 |
| 16. | APPENDIX 2: LASA SCALE | |

# **LIST OF TABLES**

| Table 1: Summary of all clinical studies of systemically administered AP | L-2 (up to September 2017) |
|---|---|
| | 23 |
| Table 2: Blood Volume during Study (up to Day 414) | 41 |

#### 1. SYNOPSIS

Protocol Number APL2-202

Official Title A Phase IIa, Open Label, Multiple Dose Study to Assess the

Safety, Efficacy and Pharmacokinetics of Subcutaneously Administered APL-2 in Subjects with Paroxysmal Nocturnal

Hemoglobinuria (PNH)

Protocol Version and Date

Version 3.0 31 January 2018

Compound APL-2

Study Phase and

Type

Phase IIa. Open-label, evidence of activity, safety, tolerability, pharmacokinetics (PK), multiple dose study.

**Study Objectives** 

The objectives of the study are to assess the safety, tolerability, efficacy and PK of multiple (SC) doses of APL-2 in subjects with paroxysmal nocturnal hemoglobinuria (PNH) who have not received treatment with eculizumab in the past.

An exploratory objective of the study is to assess the pharmacodynamics (PD) of multiple SC doses of APL-2 when administered to PNH patients.

**Study Population** 

Subjects will:

- be male and female (using contraception as specified in the protocol) and at least 18 years old
- have a diagnosis of PNH

Number of Subjects The study will be conducted alongside the ongoing Phase Ib study APL2-CP-PNH-204 (PADDOCK) to investigate APL-2 in PNH patients who have not previously received treatment with eculizumab. Safety and efficacy data from both studies will be used to support the data obtained in the Phase III confirmatory study. Up to 20 subjects will be enrolled to complete 28 days of dosing.

#### **Inclusion Criteria**

At Screening (unless otherwise specified)

- At least 18 years old (inclusive)
- Diagnosed with PNH (white blood cell (WBC) clone >10%)
- Lactose dehydrogenase (LD) ≥2 times the upper limit of normal
- Screening Ferritin ≥ normal and Total Iron Binding Capacity
   (TIBC) ≤ LLN based on central lab reference ranges. If a subject
   is receiving iron supplements at screening, the investigator must
   ensure that his/her dose has been stable for 8 weeks prior to
   enrolment and must be maintained throughout the study (see
   Section 8.4.4)
- Last transfusion within 12 months prior to screening
- Platelet count of >30,000/mm<sup>3</sup> at the screening visit
- Absolute neutrophil count >500/ mm<sup>3</sup> at the screening visit
- Women of child-bearing potential (WOCBP) must have a negative pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study
- Males must agree to use protocol defined methods of contraception and agree to refrain from donating sperm for the duration of the study
- Vaccination against Neisseria meningitides types A, C, W, Y and B, Streptococcus pneumoniae and Haemophilus influenzae Type B (Hib) either within 2 years prior to Day 1 dosing, or within 14 days after starting treatment with APL-2. Unless documented evidence exists that subjects are non-responders to vaccination as evidenced by titers or display titer levels within acceptable local limits
- Willing and able to give informed consent

#### **Exclusion Criteria**

- Prior eculizumab (Soliris®) treatment
- Active bacterial infection
- Hereditary complement deficiency
- History of bone marrow transplantation
- Concurrent severe aplastic anemia (SAA), defined as currently receiving immunosuppressive therapy for SAA including but not limited to cyclosporin A, tacrolimus, mycophenolate mofetil or anti-thymocyte globulin
- Participation in any other investigational drug trial or exposure to another investigational agent, device or procedure within 30 days

- Evidence of QTcF prolongation defined as >450 ms for males and >470 ms for females at screeningBreast-feeding women
- History of meningococcal disease

## **Endpoints**

#### **Primary Safety Endpoint:**

The primary safety endpoints of the study are the number and severity of treatment emergent adverse events (TEAEs) following administration of multiple doses of SC APL-2.

## **Primary Efficacy Endpoints:**

- Change from baseline in LD
- Change from baseline in Haptoglobin
- Change from baseline in Hemoglobin (Hb)

## Secondary Endpoints:

- APL-2 plasma concentrations (and pharmacokinetic (PK) parameters as appropriate)
- Change from baseline in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale score
- Change from baseline in reticulocyte count
- Change from baseline in total bilirubin
- Change from baseline in Linear Analog Scale Assessment (LASA) for Quality of Life
- Number of red blood cell (RBC) transfusions per month

## Exploratory PD markers include:

- Complement (CH50, AP50, and C3) levels
- C3 deposition on RBC cells
- Clonal distribution of PNH RBCs

# Planned Dose Levels

The planned dose for this single cohort study will be a daily dose of 270 mg/day however from Part 2A onwards intra-subject dose escalation up to a dose of 360 mg/day may be permitted.

The dose was determined based on cumulative safety, PK, and PD data from ongoing studies in PNH patients.

Safety data from this study will be reviewed by the SMC on a regular basis.

#### Study Design

This is a Phase IIa, open-label, multiple dose, study in patients with PNH who have not received eculizumab (Soliris®) in the past. A single cohort is planned for evaluation.

The study will be conducted alongside the ongoing Phase Ib study APL2-CP-PNH-204 (PADDOCK) to investigate APL-2 in PNH patients who have not previously received treatment with eculizumab. Safety and efficacy data from both studies will be used to support the data obtained in the Phase III confirmatory study. Up to 20 subjects will be enrolled to complete 28 days of dosing (Part 1).

Safety will be assessed throughout the study; serial blood and urine samples will be collected for these assessments. Blood samples will be collected for the assessment of APL-2 PK. Additional samples for assessment of PD will also be collected.

The study will consist of four parts:

- Part 1: subjects will receive APL-2 for 28 days.
- Part 2A: subjects may continue to receive APL-2 for a further 56 days if there is evidence of clinical benefit following review of available safety, PK and PD data by the investigator and sponsor
- Part 2B: subjects may continue to receive daily APL-2 treatment for up to 364 days if there is ongoing evidence of clinical benefit following review of the available safety, PK and PD data.
- Part 3: Safety follow up

Screening will take place within 30 days prior to the start of dosing on Day 1.

Subjects will be entered into Part 1 of the study on Day 1 at a time designated by the PI. Research nurses or other appropriately qualified research personnel will administer the SC infusions for a minimum of 3 days (Days 1-3) until the research nurse considers that the subject is both capable and confident to conduct self-administration. The subject will continue to self-administer infusions at the clinic on those days when a clinic visit occurs (Day 8, 15 and 22) and at an off-site location convenient to the subject on all other days up to Day 28 in Part 1.

Following ongoing review of available safety, PK and PD data by the investigator and sponsor, subjects showing evidence of clinical benefit may progress to Part 2A and then to Part 2B of the study and continue to receive daily doses of APL-2 until Day 84 and then until Day 364. Doses will be self-administered by the subject throughout this period at an off-site location convenient to the subject with the exception of Days 29, 36, 43, 57, 71, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 where dosing is performed by the subject at the clinical site. After the conclusion of the treatment period (Day 364), subjects will return to the clinical site for follow-up study procedures on Day 365, 379, and

393 and final study procedures at an Exit Visit on Day 414 See Study Flow Chart in Section 2.

The planned length of participation in the study for each subject is approximately 444 days (14.5 months) from Day -30 through completion of the Day 414 Exit visit procedures).

# 2. STUDY FLOW CHART

| Study Period | Part 1 – Treatment (Daily from Day 1 to Day 28) | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | | | | | | | | | | 4 | |
| Study Day | -30 | 1 | 2 | 3 | 4 to 7 | 8 | 9 to 14 | 15 | 16 to 21 | 22 | 23 to 28 |
| Informed Consent | Х | | | | | | | | | | |
| Demographics | Х | | | | | | | | | | |
| Medical, transfusion, and thrombosis history | х | | | | | | | | | | |
| Vaccination. A | | | | | | | | х | | | |
| Review entry criteria | | х | | | | | | | | | |
| Preventive antibiotic. B | | х | Х | х | х | Х | х | х | х | Х | х |
| Physical examination. C | Х | | | | | | | | | | |
| 12-lead electrocardiogram. D | Х | х | | х | | Х | | Х | | Х | |
| APL-2 administration. E | | S | S | S | Н | S | Н | S | Н | S | Н |
| Injection site assessment. F | | х | Х | х | х | Х | х | х | х | Х | х |
| Concomitant medications | Х | Х | Х | х | х | Х | х | Х | x | Х | x |
| Vital sign measurements. G | Х | Х | Х | Х | х | Х | х | Х | х | Х | x |
| Urinalysis | Х | Х | | | | х | | х | | Х | |
| Blood. I | Х | Х | | | | х | | х | | х | |
| Pharmacokinetics. I | | x (I) | Х | х | | х | | | | х | |
| Anti-APL-2 Ab assay | | х | | | | | | х | | | |
| Hematology and chemistry. | Х | х | | | | х | | х | | х | |
| Coagulation profile | Х | Х | | | | х | | х | | х | |
| Complement profile (C3, CH50 and AP50) | Х | х | | | | х | | х | | x | |
| Flow cytometry for PNH/C3 deposition | Х | х | | | | х | | х | | х | |
| Plasma Hb | Х | х | | | | х | | х | | х | |
| Pregnancy (B-human chorionic gonadotropin) | Х | | | | | | | | | | |
| Urine pregnancy test. J | | Х | | | | х | | Х | | х | |
| FACIT fatigue Scale | | Х | | | | | | Х | | | |
| LASA QoL | | х | | | | | | х | | | |
| Adverse events | | Х | Х | Х | х | Х | Х | Х | Х | Х | х |
| Thrombosis record (MAVE). K | | х | Х | х | х | Х | Х | х | Х | Х | х |

See footnotes below continuation flow chart

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

| Study Period | Part 2A - Treatment (Daily from Day 29 to Day 84) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | | 5 | | 6 | | 7 and 8 | | 9 and 10 | 11 and 12 | |
| Study Day | | <u> </u> | | | | 7 allu o | | 9 and 10 | 11 anu 12 | |
| | 29 | 30 to 35 | 36 | 37 to 42 | 43 | 44 to 56 | 57 | 58 to 70 | 71 | 72 to 84 |
| Informed Consent | | | | | | | | | | |
| Demographics | | | | | | | | | | |
| Medical, transfusion, and thrombosis history | | | | | | | | | | |
| Vaccination. A | | | | | | | | | | |
| Review entry criteria | | | | | | | | | | |
| Preventive antibiotic. B | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Physical examination. C | Х | | | | | | Х | | | |
| 12-lead electrocardiogram. D | Х | | Х | | Х | | Х | | Х | |
| APL-2 administration. E | S | Н | S | Н | S | Н | S | н | S | Н |
| Injection site assessment. F | Х | X | Х | X | Х | Х | Х | Х | Х | Х |
| Concomitant medications | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Vital sign measurements. G | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Urinalysis | Х | | Х | | Х | | Х | | Х | |
| Blood. I | Х | | Х | | Х | | Х | | Х | |
| Pharmacokinetics. I | Х | | | | Х | | | | Х | |
| Anti-APL-2 Ab assay | Х | | | | | | | | Х | |
| Hematology and chemistry. | Х | | Х | | Х | | Х | | Х | |
| Coagulation profile | Х | | Х | | Х | | Х | | Х | |
| Complement profile (C3, CH50 and AP50) | Х | | Х | | Х | | Х | | Х | |
| Flow cytometry for PNH/C3 deposition | Х | | Х | | Х | | Х | | Х | |
| Plasma Hb | Х | | Х | | Х | | Х | | Х | |
| Urine pregnancy test. J | Х | | Х | | Х | | Х | | Х | |
| FACIT fatigue Scale | Х | | | | Х | | | | Х | |
| LASA QoL | Х | | | | Х | | | | Х | |
| Adverse events | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Thrombosis record (MAVE). K | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |

See footnotes below continuation flow chart

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

| Study Period | | | | Par | t 2B - Tre | eatment (Daily | from Da | y 85 to Day 364 | 1) (L) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | 1 | 3 to 16 | 17 to 20 | | 21 to 24 | | 25 to 28 | | 29 to 32 | | 3 | 3 to 36 |
| Study Day | 85 | 86 to 112 | 113 | 114 to 140 | 141 | 142 to 168 | 169 | 170 to 196 | 197 | 198 to 224 | 225 | 226 to 252 |
| Vaccination | Х | | | | | | | | | | | |
| Preventive antibiotic. B | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Physical examination. C | Х | | | | | | | | | | | |
| 12-lead electrocardiogram. D | Х | | Х | | Х | | Х | | Х | | Х | |
| APL-2 administration. E | S | Н | S | Н | S | Н | S | Н | S | Н | S | Н |
| Injection site assessment. F | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Concomitant medications | Х | Х | Х | Х | Х | Х | Х | X | Х | Х | Х | Х |
| Vital sign measurements. G | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Urinalysis | Х | | Х | | Х | | Х | | Х | | Х | |
| Blood. I | Х | | Х | | Х | | Х | | Х | | Х | |
| Pharmacokinetics. I | Х | | Х | | Х | | Х | | Х | | Х | |
| Anti-APL-2 Ab assay | Х | | | | Х | | | | Х | | | |
| Hematology and chemistry. | Х | | Х | | Х | | Х | | Х | | Х | |
| Coagulation profile | Х | | Х | | Х | | Х | | Х | | Х | |
| Complement profile (C3, CH50 and AP50) | Х | | Х | | Х | | Х | | Х | | Х | |
| Flow cytometry for PNH/C3 deposition | Х | | Х | | Х | | Х | | Х | | Х | |
| Plasma Hb | Х | | Х | | Х | | Х | | Х | | Х | |
| Urine pregnancy test. J | Х | | Х | | Х | | Х | | Х | | Х | |
| FACIT fatigue Scale | Х | | | | Х | | | | Х | | | |
| LASA QoL Scale | Х | | | | Х | | | | Χ | | | |
| Adverse events | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Thrombosis record (MAVE) K | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | х |

See footnotes below continuation flow chart

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

| Study Period | | Part | 2B - Tre | atment (Daily f | rom Day | 85 to Day 364 | ) (L) | |
|---|---|---|---|---|---|---|---|---|
| Study Week | 3 | 37 to 40 41 to 44 | | 11 to 44 | 4 | 15 to 48 | 4 | 19 to 52 |
| Study Day | 253 | 254 to 280 | 281 | 282 to 308 | 309 | 310 to 336 | 337 | 338 to 364 |
| Informed Consent | | | | | | | | |
| Review entry criteria | | | | | | | | |
| Preventive antibiotic. B | Х | Х | Х | Х | Х | Х | Х | Х |
| Physical examination. C | Χ | | | | | | Х | |
| 12-lead electrocardiogram. D | Х | | Х | | Х | | Х | |
| APL-2 administration. E | S | н | S | н | S | н | S | н |
| Injection site assessment. F | Х | Х | Х | Х | Х | Х | Х | Х |
| Concomitant medications | Х | Х | Х | Х | Х | Х | Х | Х |
| Vital sign measurements. G | Х | Х | Х | Х | Х | Х | Х | Х |
| Urinalysis | Х | | Х | | Х | | Х | |
| Blood. I | Х | | Х | | Х | | Х | |
| Pharmacokinetics. I | Х | | Х | | Х | | Х | |
| Anti-APL-2 Ab assay | Х | | | | Х | | | |
| Hematology and chemistry. | Х | | Х | | Х | | Х | |
| Coagulation profile | Х | | Х | | Х | | Х | |
| Complement profile (C3, CH50 and AP50) | Х | | Х | | Х | | Х | |
| Flow cytometry for PNH/C3 deposition | Х | | Х | | Х | | Х | |
| Plasma Hb | Х | | Х | | Х | | Х | |
| Urine pregnancy test. J | Х | | Х | | Х | | Х | |
| FACIT fatigue Scale | Х | | | | Х | | | |
| LASA QoL Scale | Х | | | | Х | | | |
| Adverse events | Х | Х | Х | Х | Х | Х | Х | Х |
| Thrombosis record (MAVE). K | Х | Х | Х | Х | Х | Х | Х | Х |

See footnotes below continuation flow chart

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

| Study Peri | iod | Part 3 – Follow-up and Exit. (M) | | |
|---|---|---|---|---|
| Study We | eek 53 | 55 | 57 | 60 |
| Study D | <b>9ay</b> 365 | 379 | 393 | 414 |
| Informed Consent | | | | |
| Review entry criteria | | | | |
| Preventive antibiotic. B | Х | Х | | |
| Physical examination. C | Х | | | Х |
| 12-lead electrocardiogram. D | Х | | | |
| APL-2 administration. E | | | | |
| Injection site assessment. F | Х | | | |
| Concomitant medications | Х | Х | Х | Х |
| Vital sign measurements. G | Х | Х | Х | Х |
| Urinalysis | Х | Х | Х | Х |
| Blood. I | Х | Х | Х | Х |
| Pharmacokinetics. I | Х | Х | Х | Х |
| Anti-APL-2 Ab assay | Х | | | Х |
| Hematology and chemistry. | Х | Х | Х | Х |
| Coagulation profile | Х | Х | Х | Х |
| Complement profile (C3, CH50 and AP50) | х | Х | Х | Х |
| Flow cytometry for PNH/C3 deposition | Х | Х | Х | Х |
| Plasma Hb | Х | Х | Х | Х |
| Urine pregnancy test. J | Х | | Х | Х |
| FACIT fatigue Scale | Х | | Х | Х |
| LASA QoL Scale | Х | | Х | Х |
| Adverse events | Х | Х | Х | Х |
| Thrombosis record (MAVE) K | Х | Х | Х | Х |

See study flow chart footnotes on next page

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

## **FOOTNOTES:**

A. If required i.e. not previously vaccinated subjects will receive vaccinations against Neisseria meningitides types A, C, W, Y and B, Streptococcus pneumoniae and Haemophilus influenzae Type B (Hib). If the subject's first documented *Neisseria meningitidis* vaccine/s are administered at Day 15, a booster (for both vaccinations) should be administered after 2 months. If Pneumococcal vaccination is required, a dose of PCV13 will be administered at Day 15 and a dose of PPSV23 will be administered at least 8 weeks later (unless documented evidence exists that subjects are non-responders to vaccination as evidenced by titers or display titer levels within acceptable local limits). The PI will discuss with the Sponsor in regard to specific patient requirements

- B. Preventive antibiotics will be prescribed from Day 1. Antibiotics will be taken from Day 1 until 14 days after the first dose of APL-2. Specifically:
  - Day 1 to Day 14: Ciprofloxacin 500 mg twice daily (take post dose ECG before Ciprofloxacin is administered on days 1).
  - Day 15 onwards: Penicillin V 500 mg twice daily.
- C. Full physical examination will be performed at the scheduled time points indicated. A symptom-driven physical examination may be performed at other times, at the PI's discretion.
- D. If done on a dosing day, electrocardiograms (ECGs) are to be performed within 30 minutes after dosing.
- E. S = Administration at clinical site. H = Administration at subject's home, workplace, or other location convenient to the subject. Treatment may be stopped at any time if the investigator and sponsor conclude that there is no demonstration of clinical benefit to continue APL-2 administration past this point.
- F. Injection site assessment will be performed within 30 minutes after APL-2 administration. Ambulatory syringe infusion pump training will include instructions to report any injection site reaction to the PI.
- G. At clinic visits, vital signs will be measured within 2 hours prior to dosing and within 30 minutes after dosing. When APL-2 is self-administered, pre- and post-dose vital signs will not be measured.
- H. Reserved See note E.
- I. If done on a dosing day, blood samples will be taken pre-dose with the exception that on Day 1 only a pharmacokinetic sample will be taken pre-dose and at a minimum of 2.5 hours post-dose or immediately prior to discharge from the clinic (if subject is kept at the clinic longer than 2.5 hours).
- J. If done on a dosing day, urine pregnancy test should be completed for WOCBP prior to dosing.
- K. MAVE = Major Adverse Vascular Event. Ambulatory syringe infusion pump training will include instructions to report any events to the PI.
- L. If dose is increased during Part 2B, subjects will come back to the clinical site for safety visits every other week for the first 6 weeks of the dose change. These visits may alternate with the monthly visits and should be recorded as unscheduled visits. The same procedures listed under the monthly visits will be performed.
- M. Subjects that discontinue dosing at any time during Part 1, 2A or 2B will move directly into Part 3 for safety follow up visits.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

# 3. ABBREVIATIONS

| ADA | Anti-drug Antibodies |
|-------|----------------------------------------------------|
| ADL | Activities of daily living |
| AE | Adverse event |
| ALP | Alkaline phosphatase |
| ALT | Alanine aminotransferase |
| AP50 | Alternative Pathway |
| aPTT | Activated partial thromboplastin time |
| AST | Aspartate aminotransferase |
| BID | Twice Daily |
| BUN | Blood urea nitrogen |
| °C | Degrees Celsius |
| C3 | Complement Component 3 |
| CD71+ | Transferrin Receptor |
| CK | Creatine kinase |
| cm | Centimeter |
| CRF | Case report form |
| CS | Clinically significant abnormality |
| ECG | Electrocardiogram |
| FACIT | Functional Assessment of Chronic Illness Therapy |
| FDA | Unites States Foods and Drug Administration |
| g | Gram(s) |
| GCP | Good clinical practice |
| GGT | Gamma-glutamyl transpeptidase |
| GLP | Good laboratory practice |
| μg | Microgram(s) |
| Hb | Haemoglobin |
| hERG | Human ether-à-go-go-related gene |
| Hib | Haemophilus influenzae Type B (vaccine) |
| IB | Investigator's brochure |
| ICH | International Conference on Harmonization |
| IEC | Institutional Ethics Committee |
| IRB | Institutional Review Board |
| ITT | Intent-to-Treat |
| IV | Intravenous |
| IVT | Intravitreal |
| kDa | Kilodalton |
| kg | Kilogram(s) |
| L | Litre(s) |
| LASA | Linear Analog Scale Assessment for Quality of Life |
| LD | Lactate dehydrogenase |

| LLN | Lower Limit of Normal |
|------------------|-------------------------------------------------------|
| MAC | Membrane attack complex |
| MAVE | Major Adverse Vascular Event |
| MedDRA® | Medical Dictionary for Regulatory Activities |
| mg | Milligram(s) |
| mL | Millilitre(s) |
| MOP | Manual of Procedures |
| NCS | Not clinically significant |
| NOEL | No observed effect level |
| NOAEL | No observed adverse effect level |
| NZW | New Zealand White |
| PCV13 | Pneumococcal conjugate vaccine |
| PD | Pharmacodynamic(s) |
| PEG | Polyethylene glycol |
| PEG40 | Polyethylene glycol (40 kDa nominal molecular weight) |
| PI | Principal Investigator or designee |
| PK | Pharmacokinetic(s) |
| PPSV23 | Pneumococcal polysaccharide vaccine 23 |
| PT | Prothrombin time |
| PNH | Paroxysmal nocturnal hemoglobinuria |
| QTc | Corrected QT interval |
| QTcB | Bazett's correction |
| QTcF | Fridericia's correction |
| RBC | Red blood cell |
| SAA | Severe aplastic anaemia |
| SAE | Serious adverse event |
| SAP | Statistical Analysis Plan |
| SC | Subcutaneous |
| SMC | Safety Monitoring Committee |
| SOP | Standard operating procedure |
| t <sub>1/2</sub> | Serum half-life |
| TEAE | Treatment-emergent adverse event |
| TK | Toxicokinetic(s) |
| ULN | Upper Limit of Normal |
| WBC | White blood cell |
| WHO | World Health Organization |
| WOCBP | Woman of Child-Bearing Potential |

## 4. INTRODUCTION

# 4.1 Background

This study is being conducted as part of a series of studies for the clinical development of APL-2. The study will be conducted in compliance with the protocol, Good Clinical Practice (GCP), and

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

applicable regulatory requirements. The subject population will be comprised of adult male and female subjects with paroxysmal nocturnal hemoglobinuria (PNH).

## 4.1.1 Paroxysmal Nocturnal Hemoglobinuria

PNH is an acquired, clonal, non-malignant hematological disease characterized by complement-mediated RBC hemolysis with or without hemoglobinuria, an increased susceptibility to thrombotic episodes, and/or some degree of bone marrow dysfunction. The onset of PNH is often insidious. Although there have been reports of spontaneous remission, the course of the disease is generally chronic and progressive.

It has been known for many years that PNH is caused by complement-mediated lysis of erythrocyte clones lacking functional CD55 and CD59 on their surface to protect them against this process. As such, these erythrocytes are particularly susceptible to the membrane attack complex (MAC) and have been shown to lyse readily in the presence of complement activation.

Any therapy that effectively inhibits MAC formation is anticipated to be a plausible candidate-treatment for PNH. Indeed, eculizumab is a monoclonal anti-C5 antibody that inhibits the formation of the MAC, and eculizumab treatment has been approved for the treatment of this serious condition. However, inhibition of MAC formation does not appear to be sufficient to fully control the disease, as many PNH patients receiving eculizumab treatment still suffer from anemia, with only roughly 13% of patients being classified as complete responders, i.e. achieving transfusion independence and normal Hb levels. Most of the patients (53%) were classified as partial responders with decreased transfusion needs and reduced LD, and 33% of patients were poor responders, with unchanged transfusion needs and persistent symptoms (DeZern, 2013).

Recent studies have suggested that significant opsonization of PNH erythrocytes by C3 fragments is observed in patients receiving eculizumab treatment. This opsonization is believed to cause the removal of erythrocytes by the spleen and the liver, resulting in extravascular hemolysis. Extravascular hemolysis can be significant in a subset of eculizumab-treated PNH patients and is considered to be the principal contributor to the lack of complete eculizumab response in most patients. It is reasonable, therefore, to expect that a treatment able to inhibit both MAC formation and C3 opsonization will provide improved therapeutic benefit to PNH patients compared to eculizumab.

An overview of available information regarding APL-2 follows below. Further details can be found in the APL-2 Investigator's Brochure (Apellis Pharmaceuticals, June 2017).

#### 4.1.2 APL-2

APL-2 is formed by a pentadecapeptide (combining a cyclic tridecapeptide active C3-inhibiting moiety and a 2-amino acid linker) covalently coupled to each end of a linear 40 kDa PEG chain, so there are two peptide moieties per molecule of APL-2.

The peptide portion of the drug binds to complement C3 and is a broad inhibitor of the complement cascade, a biological process that is part of innate immunity and is involved in multiple inflammatory processes. The PEGylation of the molecule imparts slower elimination from mammalian systems following administration.

APL-2 injection (drug product) is a solution of APL-2 in 5% dextrose or a solution of APL-2 in acetate-buffered mannitol or a solution of APL-2 in acetate-buffered sorbitol for SC administration. APL-2 is being developed for the treatment of paroxysmal nocturnal hemoglobinuria (PNH).

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

#### 4.1.3 Nonclinical Data

## 4.1.3.1 Pharmacology

Primary Pharmacology: Subcutaneous (SC) and intravenous (IV) doses of APL-2 were shown to be pharmacologically active (as measured by a drop in CH50) in monkeys as soon as 8 hours following initial administration and persisting up to 72 hours after the last dose. *Ex vivo* studies conducted with blood from PNH patients revealed that an APL-2 concentration of ≥100 μg/mL can protect PNH erythrocytes (RBCs) from complement-mediated lysis while simultaneously preventing RBC opsonization by C3 fragments. APL-2 was as effective as eculizumab, an anti-C5 monoclonal antibody approved for PNH, in protecting PNH erythrocytes against membrane attack complex-mediated hemolysis but, unlike eculizumab, APL-2 was also effective in preventing opsonization of those cells by C3 fragments.

**Safety Pharmacology:** The potential for APL-2 to inhibit human ether-a-go-go gene (hERG)-encoded ion channels and pose a risk for cardiac arrhythmias indicates that such a risk is low. Similarly, no evidence of APL-2-related adverse effects on myocardial conduction, cardiovascular and respiratory systems, and body temperature control mechanisms have been observed in either rabbits or monkeys.

## 4.1.3.2 Pharmacokinetics

Pharmacokinetic (PK) and toxicokinetic (TK) assessments of APL-2 have been investigated after IV and SC administration to New Zealand White (NZW) rabbits and cynomolgus monkeys. The PK behavior of APL-2 in rabbits and monkeys has been consistent with the expected PK behavior of a PEGylated peptide. APL-2 is readily absorbed from SC injections in both species, with an estimated bioavailability of approximately 85% in monkeys. Repeated administrations of APL-2 have indicated that absorption is non-linear at higher doses, and the potential for bioaccumulation exists. No gender-related differences have been observed in either species after 6 or 9 months of SC dosing in rabbits and monkeys, respectively. Terminal elimination half-lives (t<sub>1/2</sub>), estimated during 4-week, drug-free, recovery phases of the 28-day SC studies were between 2.48–2.78 days in rabbits and 6.29–8.25 days in monkeys. Similarly, the t<sub>1/2</sub> was estimated to be between 2.3 and 2.6 days in rabbits and 6.0 days in monkeys after two IV doses separated by 14 days.

## 4.1.3.3 Toxicology

The toxicological potential of APL-2 has been investigated in repeat-dose toxicity studies in rabbits and monkeys across three routes of administration (SC, IV, IVT) under a testing strategy designed to facilitate differentiation between potential changes attributable to APL-2 per se and those attributable to the PEG40 domain of the drug molecule.

Daily subcutaneous administration of APL-2 and PEG40 for a duration of 6 months in rabbits and 9 months in monkey were associated with little systemic toxicity noted in either species beyond observations in the kidney (noted below). APL-2 and PEG40 were weakly to mildly immunogenic in rabbits, but not significantly immunogenic in monkeys. Single- or multi-tissue (or multi-organ) macrophage vacuolation was consistently observed in both species, and generally comparable in incidence and severity between APL-2- and PEG40-treated groups; thus, it was concluded the finding were caused by the PEG40 domain present within APL-2. Renal tubular degeneration was observed with a higher incidence in the monkey 9-month study in APL-2-treated animals compared to the PEG40-treated ones and was concluded to be APL-2 related.

The no-observed-adverse-effect-level (NOAEL) for SC-administered APL-2 was <1 mg/kg/d in rabbits and approximately 7 mg/kg/d in monkeys after 6- and 9-month chronic dosing, respectively.

Intravenous arms included in the 28-day repeat-dose SC studies of APL-2 in rabbits and monkeys suggested that IV-administered APL-2 was well-tolerated in both species, with only vacuolation of

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

tubular epithelial cells in the kidney observed microscopically in rabbits (which, again, was deemed to be caused in part by the PEG40 domain of APL-2). IV APL-2 was mildly immunogenic in rabbits (albeit less than what was observed by the SC route), and without immunologic effects in monkeys. The no-observed-effect-level (NOEL) by the IV route of administration for both rabbits and monkeys was determined to be ≥42 mg/kg after two doses separated by 14 days.

Repeated intravitreal administration (i.e. once every 4 weeks) of APL-2 to monkeys for up to 9 months was well-tolerated and revealed no drug-related systemic or ophthalmological changes. APL-2 may be minimally immunogenic when administered intravitreally, as evidenced by a single monkey having a marginal titer of APL-2 antibodies. The NOEL by the IVT route of administration for monkeys was determined to be ≥24.8 mg/eye.

APL-2 has not demonstrated genotoxic potential in any *in vitro* or *in vivo* genotoxicity assays conducted, to date.

#### 4.1.4 Clinical Data

To date, two Phase I studies in healthy volunteers have been conducted in order to assess safety and PK parameters of APL-2 administered as single and multiple dose SC injections and to guide dose selection for clinical studies in PNH subjects.

A single Phase I single ascending dose study has evaluated intravenous dosing of APL-2 in healthy volunteers.

A further five Phase I studies evaluating APL-2 delivered by SC injection are either planned or ongoing. These include two studies in healthy volunteers, a study in subjects with severe renal impairment and two ongoing clinical studies in PNH patients.

A phase IIa study in patients with autoimmune hemolytic anemia is also ongoing.

Table 1 summarises the information for all completed and ongoing studies evaluating systemic administration of APL-2.

Table 1: Summary of all clinical studies of systemically administered APL-2 (up to September 2017)

| Protocol<br>Number<br>/Phase/Status | Protocol Title | Study Population<br>Subjects<br>Planned/Treated | Endpoints | Planned Dosage Regimen |
|---|---|---|---|---|
| SUBCUTANEOUS | | | | |
| APL-CP0713-1<br>Phase I<br>Complete | Phase I, Double-blind,<br>Randomized, Single<br>Ascending Dose Study in<br>Healthy Volunteers | 31 healthy<br>volunteers<br>APL-2: 24/24<br>Placebo: 7/7 | Safety, tolerability,<br>PK and PD of<br>single ascending<br>doses (SAD) of<br>APL-2 | SAD: 45, 90, 180, 360, 720, 1440 mg<br>Single dose |
| APL-CP1014<br>Phase I<br>Complete | Phase I, Double-blind,<br>Randomized, Multiple<br>Ascending Dose Study in<br>Healthy Volunteers | 20 healthy<br>volunteers<br>APL-2: 16/6<br>Placebo: 4/4 | Safety, tolerability,<br>PK and PD of<br>multiple ascending<br>(MAD) doses of<br>APL-2 | MAD: 30, 90, 180, 270 mg/day for 28 days |
| APL2-CP-PV-<br>205<br>Phase I<br>Ongoing | A Phase I, Single-Dose,<br>Open-Label Study to Evaluate<br>the Effect of Renal Impairment<br>on the Pharmacokinetics of<br>APL-2 | 8 subjects with<br>severe renal<br>impairment and 8<br>matched controls<br>APL-2: 16/1 | Comparative PK<br>between subjects<br>with severe renal<br>impairment and<br>matched controls | 270 mg single dose |
| APL2-101<br>Phase I<br>Ongoing | A Phase I, Double-Blind,<br>Randomized Study of Daily,<br>Twice-Weekly and Once-<br>Weekly APL-2 in Healthy<br>Volunteers | 22 Healthy<br>Volunteers<br>APL-2: 16/0<br>Placebo: 6/0 | Safety, tolerability,<br>PK and PD of APL-<br>2 | 360 mg daily<br>1300 mg twice weekly<br>2600 mg weekly |

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

| Protocol<br>Number<br>/Phase/Status | Protocol Title | Study Population<br>Subjects<br>Planned/Treated | Endpoints | Planned Dosage Regimen |
|---|---|---|---|---|
| | | | | TBD (Final Cohort if dosed) |
| APL-2-102<br>Phase I<br>Ongoing | Phase I, Double-blind,<br>Randomized, Single<br>Ascending Dose Study in<br>Healthy Japanese Volunteers | 20 Healthy<br>Volunteers<br>APL-2: 16/0<br>Placebo: 4/0 | Safety, tolerability,<br>PK and PD of<br>single ascending<br>doses (SAD) of<br>APL-2 | SAD: 180, 360, 720, 1440 mg Single dose |
| APL-CP0514<br>Phase I<br>Ongoing | An Open Label, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of APL-2 as an Add-On to Standard of Care in Subjects with PNH. | 12 patients with<br>PNH – Eculizumab<br>APL-2: 12/12 <sup>1</sup> | Safety, tolerability,<br>PK and PD | Cohort 1: 25 mg SD followed by 28 days washout then 5 mg/day for 28 days Cohort 2: 50 mg SD followed by 28-day washout then 30 mg/day for 28 days Cohort 3: 180 mg/day for 28 days Cohort 4: 270 mg/day for up to 2 years (ongoing) |
| APL2-CP-PNH-<br>204<br>Phase Ib<br>Ongoing | A Phase Ib, Open Label, Multiple Ascending Dose, Pilot Study to Assess the Safety, Preliminary Efficacy and Pharmacokinetics of Subcutaneously Administered APL-2 in Subjects with PNH. – PADDOCK – | 9 patients with PNH - Eculizumab naïve APL-2: 9/6 <sup>2</sup> | Safety, tolerability,<br>PK and PD | Cohort 1: 180 mg/day for 28 days <sup>3</sup> Cohort 2: 270 mg/day for up to 365 days (ongoing) |
| APL2-CP-AIHA-<br>208<br>Phase IIa<br>Ongoing | An Open Label, Prospective<br>Study to Assess the Safety,<br>Tolerability, Efficacy and<br>Pharmacokinetics of APL-2 in<br>Subjects with Warm Antibody<br>Autoimmune Hemolytic<br>Anemia (wAIHA) or Cold<br>Agglutinin Disease (CAD) | 6 patients with<br>wAIHA and 6<br>patients with CAD<br>APL-2: 12/0 | Safety, tolerability,<br>PK and PD of SAD<br>APL-2 | 270 mg/day for 1 year<br>360 mg/day for 1 year |
| INTRAVENOUS | | | | |
| APL2-CP-HV-<br>401<br>Phase I<br>Complete | A Phase I, Double-blind,<br>Randomized, Placebo-<br>Controlled, Single Ascending<br>Dose Study of Intravenous<br>APL-2 in Healthy Volunteers | 20 healthy<br>volunteers<br>APL-2: 16/16<br>Placebo: 4/4 | Safety, tolerability,<br>PK and PD of SAD<br>APL-2 | SAD: 200, 600, 1500 and 2300 mg IV - Single dose |

# 4.1.5 Completed Clinical Studies in Healthy Volunteers

The two completed clinical studies investigating the safety, tolerability and PK of single (APL-CP-0713-1) and multiple (APL-CP-1014) SC doses of APL-2 in healthy volunteers showed that overall, single doses of APL-2, up to a dose of 1440 mg, and repeated daily doses of APL-2 up to a dose of 270 mg, appeared safe and well tolerated when administered to healthy volunteers by SC injection.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

<sup>&</sup>lt;sup>1</sup> One subject is included in 3 cohorts and is counted three times and one subject is included in two cohorts and is counted twice.

<sup>&</sup>lt;sup>2</sup> One subject is included in 2 cohorts and is counted twice.

<sup>&</sup>lt;sup>3</sup> One subject received only a single dose of 180 mg then withdrew consent.

Serum APL-2 concentrations generally increased linearly with dose. APL-2 was slowly absorbed into the systemic circulation with median  $T_{\text{max}}$  values between 4.5 and 6 days across the dose groups. APL-2 serum concentration declined in a steady mono-exponential manner with a consistent rate of decay across two studies for all dose groups. Both studies demonstrated a slow terminal elimination with median  $t\frac{1}{2}$  values between 8 and 10 days.

Plasma complement C3 increased with increasing dose and a general dose-dependent reduction in AP50 was observed following multiple dosing with APL-2. Pharmacodynamic (PD) observations were consistent with a conclusion that APL-2 interacts with complement C3 and inhibits its activation.

Further details can be found in the current APL-2 Investigator's Brochure.

## 4.1.6 Ongoing Clinical Studies

As of September 2017 there were two ongoing Phase I clinical studies evaluating SC administered APL-2 in PNH patients (APL-CP0514 and APL-2-CP-PNH-204). An interim analysis has been performed for both studies with a data cut at 85 days of treatment for all subjects:

- 1. APL-2-CP-PNH-204 is a Phase Ib, open-label study in patients with PNH who are not receiving eculizumab. The study is comprised of 2 cohorts with three subjects in cohort 1 (180 mg/day APL-2) and at least 6 subjects in Cohort 2 (270 mg/day APL-2). Cohort 1 has completed and Cohort 2 is ongoing. Two of 3 subjects who have entered into Cohort 2 have completed 3 months of treatment with APL-2 270 mg/day. The third subject withdrew, for personal reasons, after receiving 29 days of treatment. A protocol amendment allowed intra-subject dose escalations up to 360 mg/day. Based on the clinical benefit observed, both subjects who continued dosing beyond 29 days were eligible to enter an extension phase (Part 2B) allowing them to continue to receive dosing with APL-2 for up to 1-year. One subject withdrew for personal reasons; 1 subject entered the extension phase and received daily doses of APL-2 for >8 months including doses of 360 mg for >3 months, but was diagnosed with a malignancy, unrelated to the study drug, and treatment was withdrawn in April 2017; the remaining subject continues to receive APL-2 270 mg/day. Based on the emerging data, a country specific protocol was submitted and the subject may continue dosing for up to 729 days. This study is currently being expanded into Asia.
- 2. APL-CP0514 is a Phase Ib, open-label study being conducted at multiple clinical sites in the United States to assess the safety, tolerability, PK and PD of APL-2 as an add-on to eculizumab in subjects with PNH. The study is comprised of 4 cohorts in total; 3 cohorts (Cohorts 1-3) with two subjects per cohort, and one cohort with six subjects (Cohort 4). Cohorts 1 to 3 have completed and Cohort 4 is ongoing. All six subjects in Cohort 4 completed at least 3 months of treatment with APL-2 270 mg/day. A protocol amendment allowed intra-subject dose escalations up to 360 mg/day. Based on the clinical benefit observed all subjects entered an extension phase allowing them to continue to receive dosing with APL-2 for up to 1 year. Two subjects have withdrawn from the study; 1 subject became pregnant and was withdrawn as per protocol and the 2<sup>nd</sup> subject was withdrawn following a number of adverse events related to other co-morbidities. Based on the emerging data, dosing will continue for up to 729 days.

Across the two studies in PNH patients, a total of 14 subjects with PNH have been dosed with APL-2, with 9 having received 270 mg/day for 28 day and 8 having received ≥270 mg/day for >3 months including 2 who have received 360 mg/day for 2 months. APL-2 has been generally well tolerated in these subjects. At approximately bi-monthly intervals, all safety data from each study is reviewed by members of an independent SMC who are responsible for providing recommendations with respect to monitoring and continuation of the studies.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

As of the 1<sup>st</sup> September 2017, there have been a total of seventeen SAEs reported in five out of fourteen subjects across the two studies. Of these, fourteen are considered to be unrelated/unlikely to APL-2 and three have been assigned a causality of 'possibly related' to APL-2 by the Sponsor. Those that are considered possibly related include hypersensitivity reaction, and two incidences of increased ALT in a single subject with a history of hepatobiliary disease and similar ALT increases prior to study entry.

Overall, SC administration of APL-2 in PNH patients in the two ongoing clinical studies has been generally safe and well tolerated.

#### 4.2 Rationale

## 4.2.1 Purpose of the Study

This study will investigate APL-2 in patients with PNH that have not received treatment with eculizumab in the past. The assessments of safety, tolerability, preliminary efficacy, PK, and PD following administration of multiples doses of APL-2 will be added to the data generated in study APL2-CP-PNH-204 to help guide decisions to further develop the drug.

#### 4.2.2 Dose Selection

The toxicological data accumulated from the animal studies were used to guide dose selection during the Phase I single ascending dose and multiple ascending dose studies in HVs (protocols APL-CP0713-1 and APL-CP1014 respectively). In particular, the highest doses were selected based on exposure predicted by the PK model and compared with the exposures measured at the no observed adverse effect level (NOAEL) in monkeys.

The planned dose of APL-2 is 270 mg/d. Dose selection was based on targeting a level of complement C3 inhibition that will not reduce the levels of uncomplexed C3 (or free C3) to no less than about ~10 % of the normal levels of C3 (approximately 1.0-1.3 g/L). The rationale for this limit was to preserve some level of complement activity required for adequate immune function. Using a Target Mediated Drug Disposition (TMDD) PKPD model (Magar, 2001) the relationship between APL-2 PK concentration and complement C3 binding has been well characterized. Subsequently, model predictions have been derived to investigate the APL-2 dose-response. Using this TMDD PKPD model, the predicted level of free C3 at the dose of 270 mg/d was calculated to be approximately 0.13 g/L. For comparison, at the higher dose of 360 mg/d the predicted level of free C3 is approximately 0.08 g/L, which is slightly below the self-determined limit of 0.1-0.13 g/L.

Dose selection is further supported by emerging clinical data from PNH patients receiving daily doses of SC APL-2. To date, no safety issues have emerged that preclude further clinical investigation with the 270 mg/d dose.

The proposed dose of 270 mg/d should not produce a significant increase in exposure when compared to the previous human experience of a bolus injection of 270 mg/d and is supported by the 28-day repeat dose toxicology study in cynomolgus monkeys (study 13CATX-004) and human PK data derived from the single- and multiple-dose ascending studies in healthy volunteers (protocols APL-CP0713-1 and APL-CP1014).

## 4.3 Risk/Benefit

A number of safety monitoring practices are required by this protocol (i.e. physical examination, vital signs, 12-lead ECG, hematology, serum chemistry, urinalysis, coagulation, prompt reporting of pre-defined AEs of special interest, and AE questioning) in order to protect the subjects' safety.

Injection/infusion site and pump use safety will be assessed during clinical visits, and any significant finding from the assessment will be reported as an AE (see Section 11).

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

The volume of blood planned for collection from each subject over the course of the study (see Section 10.6) will be minimized, in order to minimize the impact on the overall health of these anemic subjects. If dose is increased during part 2B, additional blood draws will be required.

Systemic complement inhibition might predispose individuals to infections caused by encapsulated organisms, including *Streptococcus pneumoniae*, *Neisseria meningitides*, and *Haemophilus influenzae*. Prophylactic antibiotic therapy (ciprofloxacin 500 mg BID) will be prescribed to all subjects from Day 1 (commencing after first administration of APL-2 and the subsequent post-dose PK sample and ECG) to Day 14. At Day 15 all subjects will discontinue treatment with ciprofloxacin and receive vaccinations, if required, against *Streptococcus pneumoniae*, *Neisseria meningitides A, C, W, Y and B*, and *Haemophilus influenza*. Prophylactic antibiotic therapy (penicillin V 500 mg twice a day) will be prescribed to all subjects from Day 15 and will be taken by subjects until 14 days after the final dose of APL-2 to minimize potential infection risk. Body temperature and vital signs will be monitored periodically and relevant blood parameters monitored regularly throughout the study to assess for signs of infection. The principal investigator (PI) should be contacted immediately in the event of a suspected infection despite prophylactic antibiotic treatment for guidance and appropriate action to be taken.

Serious and occasionally fatal hypersensitivity (anaphylactic) reactions have been reported in patients on beta-lactam antibiotic (e.g. penicillin, amoxicillin, etc.) therapy. These reactions are more likely to occur in individuals with a history of penicillin hypersensitivity. Before initiating therapy with penicillin V, careful inquiry should be made concerning previous hypersensitivity reactions to penicillins or cephalosporins. Patients with a known hypersensitivity to penicillin/amoxicillin may be prescribed erythromycin 500 mg twice daily or Azithromycin 500 mg 3 times per week as alternative treatments at the outset as an alternative treatment at the outset (see Section 8.4 for details).

Other frequently reported adverse effects in patients taking penicillin are diarrhea/loose stools, nausea, skin rashes, urticaria and vomiting. Patients should, therefore, be advised that these reactions may occur. Treatment may be switched to erythromycin 500 mg twice daily or Azithromycin 500 mg 3 times per week (see Section 8.4 for details) if there is evidence of penicillin-related intolerability (such as nausea and diarrhea).

There is an anticipated health benefit for trial participants from receipt of study drug. At the proposed dose levels of APL-2, a significant decrease in complement-mediated hemolytic activity was observed in all APL-2-treated subjects (both treatment-naïve and treated previously with eculizumab) in PNH Phase Ib studies and in HV studies. APL-2 is therefore expected to reduce complement-mediated hemolytic activity in PNH patients. In this context, a careful evaluation of the risk/benefit ratio should be made. APL-2 at the proposed doses has been deemed safe for up to 9 months of administration in preclinical and 28 days in healthy volunteer studies. In addition, in both studies in subjects with PNH (See Section 4.1.4), ongoing treatment with APL-2 270 mg/day has been well-tolerated and has provided clinical benefit to subjects either alone or as an add-on to eculizumab. Based on this data we propose to continue to administer APL-2 to PNH patients for up to 364 days (1 year). See Planned Dose Levels and Dosing Schedule in Section 8.3.2.

If efficacious and safe, APL-2 is expected to continue to improve Hb levels and reduce transfusion dependency in these subjects throughout the treatment period of 364 days. Subjects will be assessed by the Investigator every month for Part 2A and Part 2B. The available safety, PK and PD data will be reviewed by the Investigator and Sponsor on an ongoing basis. If the dose of APL-2 is increased to above 270 mg/day, the subject will be assessed by the investigator every 2 weeks (recorded as unscheduled visits) for the first 6 weeks after the dose increase, subjects will then revert to appropriate time intervals for site visits according to the protocol schedule. APL-2 will only be continued in the absence of any safety concerns and with evidence of clinical benefit to the subject, as determined by the Investigator and the Sponsor.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

If a benefit is observed an extension study will be considered and will be submitted as a further protocol amendment or as a follow-up study.

#### 5. STUDY OBJECTIVES AND ENDPOINTS

## 5.1 Study Objectives

The objectives of the study are to assess safety, tolerability, preliminary efficacy and PK of multiple SC doses of APL-2 in subjects with paroxysmal nocturnal hemoglobinuria (PNH) who have not received treatment with eculizumab (Soliris)® in the past.

An exploratory objective of the study is to assess the pharmacodynamics (PD) of multiple SC doses of APL-2 when administered to PNH subjects. See "Study Endpoints" in Section 5.2.

# 5.2 Study Endpoints

#### Primary Safety Endpoint:

The primary safety endpoints of the study are the number and severity of treatment emergent adverse events (TEAEs) following administration of multiple doses of SC APL-2.

## **Primary Efficacy Endpoints:**

- Change from baseline in LD
- Change from baseline in Haptoglobin
- Change from baseline in Hb

#### Secondary Endpoints:

- APL-2 plasma concentrations (and PK parameters as appropriate)
- Change from baseline in FACIT Fatigue Scale score
- Change from baseline in reticulocyte count
- Change from baseline in total bilirubin
- Number of RBC transfusions per month
- Change from baseline in Linear Analog Scale Assessment (LASA) for Quality of Life

## **Exploratory PD markers include:**

- Complement (CH50, AP50, and C3) levels
- C3 deposition on RBC cells
- Clonal distribution of PNH RBCs

#### 6. STUDY DESIGN

This is a Phase IIa, open-label, multiple dose, study in patients with PNH who have not received eculizumab (Soliris®) in the past. A single cohort of subjects is planned for evaluation.

Safety will be assessed throughout the study; serial blood and urine samples will be collected for these assessments. Blood samples will be collected for the assessment of APL-2 PK. Additional samples for assessment of PD will also be collected.

The study will consist of four parts;

Part 1: Subjects will receive APL-2 for 28 days.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

- Part 2A: Following review of available safety, PK and PD data by the investigator and sponsor, subjects showing evidence of clinical benefit may progress to Part 2A of the study and continue to receive daily doses of APL 2 until Day 84.
- Part 2B: Following review of available safety, PK and PD data by the investigator and sponsor subjects showing evidence of clinical benefit may progress to Part 2B of the study and continue to receive daily doses of APL 2 until Day 364.
- Part 3: Safety follow up

Screening will take place within 30 days prior to the start of dosing on Day 1.

Subjects will be entered into Part 1 of the study on Day 1 at a time designated by the PI. Research nurses or other appropriately qualified research personnel will administer the SC infusions for a minimum of 3 days (Days 1-3) until the research nurse considers that the subject is both capable and confident to conduct self- administration. The subject will continue to self-administer infusions at the clinic on those days when a clinic visit occurs (Day 8, 15 and 22) and at an off-site location convenient to the subject on all other days up to Day 28 in Part 1. Following review of available safety, PK and PD data by the investigator and sponsor subjects demonstrating clinical benefit from the treatment may progress to Part 2A of the study and continue to receive daily doses of APL-2 until Day 84, and then may progress to Part 2B of the study and continue to receive daily doses of APL-2 until Day 364. Doses will be self-administered throughout this period at an off-site location convenient to the subject with the exception of Days 29, 36, 43, 57, 71, 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 where dosing is performed by the subject at the clinical site. If a subject has a sub-optimal clinical response during daily dosing with 270 mg APL-2, the dose may be increased up to 360 mg/day during part 2A, and doses will be administered at the clinical site every 2 weeks for the first 6 weeks after commencing the higher dose. After the conclusion of the treatment period (Day 364), subjects will enter Part 3 of the study and return to the clinical site for follow-up study procedures on Day 365, 379, and 393 and final study procedures at an Exit Visit on Day 414. See Study Flowchart in Section 2.

The planned length of participation in the study for each subject is approximately 444 days (from Day –30 through completion of the Day 414 Exit visit procedures). Interim PK and PD analyses may be performed to reconsider the sampling time points as the study progresses.

An independent Safety Monitoring Committee (SMC) will assess the progress and cumulative safety/tolerability data of the study on a regular basis.

## **Continuation of treatment – Decision scheme**



## 7. SUBJECT SELECTION

The study will be conducted alongside the ongoing Phase Ib study APL2-CP-PNH-204 (PADDOCK) to investigate APL-2 in PNH patients who have not previously received treatment with eculizumab. Safety and efficacy data from both studies will be used to support the data obtained in the Phase III confirmatory study. Up to 20 subjects will be enrolled to complete 28 days of dosing.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

#### 7.1 Inclusion Criteria

At Screening (unless otherwise specified), subjects must fulfill all of the following inclusion criteria to be eligible for participation in the study:

- 1. At least 18 years old (inclusive)
- 2. Diagnosed with PNH (WBC clone >10%)
- 3. Lactose dehydrogenase ≥2 times the upper limit of normal
- 4. Screening Ferritin ≥ normal and Total Iron Binding Capacity (TIBC) ≤ LLN based on central lab reference ranges. If a subject is receiving iron supplements at screening, the investigator must ensure that his/her dose has been stable for 8 weeks prior to enrolment and must be maintained throughout the study (see Section 8.4.4)
- 5. Last transfusion within 12 months prior to screening
- 6. Platelet count of >30,000/mm<sup>3</sup> at the screening visit
- 7. Absolute neutrophil count >500/ mm<sup>3</sup> at the screening visit
- 8. Women of child-bearing potential (WOCBP) must have a negative pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study
- 9. Males must agree to use protocol defined methods of contraception and agree to refrain from donating sperm for the duration of the study
- 10. Vaccination against Neisseria meningitides types A, C, W, Y and B, Streptococcus pneumoniae and Haemophilus influenzae Type B (Hib) either within 2 years prior to Day 1 dosing, or within 14 days after starting treatment with APL-2. Unless documented evidence exists that subjects are non-responders to vaccination as evidenced by titers or display titer levels within acceptable local limits
- 11. Willing and able to give informed consent

#### 7.1.1 Approved methods of contraception

Approved methods of contraception include: oral contraceptives, intrauterine device, medically acceptable barrier methods (diaphragm or condom), implantable or injectable contraceptives (like Norplant or DepoProvera) or removable birth control device (like NuvaRing or Evra patches); and/or surgical sterilization (at least 6 months before dosing). Subjects practicing abstinence and coitus interruptus (pull out method) must agree to use an approved method of contraception during the study.

#### 7.2 Exclusion Criteria

Subjects will be excluded from the study if there is evidence of any of the following criteria at screening or check-in, as appropriate.

- 1. Prior eculizumab (Soliris®) treatment
- 2. Active bacterial infection
- 3. Hereditary complement deficiency
- 4. History of bone marrow transplantation
- Concurrent SAA, defined as currently receiving immunosuppressive therapy for SAA including but not limited to cyclosporin A, tacrolimus, mycophenolate mofetil or antithymocyte globulin

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

- 6. Participation in any other investigational drug trial or exposure to other investigational agent, device or procedure within 30 days
- 7. Evidence of QTcF prolongation defined as >450 ms for males and >470 ms for females at screening
- 8. Breast-feeding women
- 9. History of meningococcal disease

#### 8. STUDY TREATMENTS

#### 8.1 Allocation to Treatment

Each subject will be assigned a unique identification number upon screening. Subjects who complete the study screening assessments and meet all the eligibility criteria will be scheduled to enter the study and receive study treatment.

## 8.2 Blinding

None; this is an open-label study.

#### 8.3 Treatments Administered

Sterile solutions of APL-2 up to 40 mg/mL in acetate-buffered mannitol administered by Subcutanoues infusion.

## 8.3.1 Drug supplies

# 8.3.1.1 Identity of Investigational Products

APL-2 will be supplied as a sterile solution of APL-2 in acetate-buffered mannitol at concentrations of up to 40 mg/mL, supplied in stoppered glass vials.

#### 8.3.1.2 Study Supplies

The Sponsor will supply sufficient quantities of APL-2 drug product to allow completion of this study. The lot numbers, manufacture dates, and expiration dates of the drugs supplied will be recorded in the final report. The Sponsor will also supply needles, syringes, and ambulatory syringe infusion pumps as required. Refer to the Study Operations Manual for further information.

APL-2 acetate-buffered mannitol solution should be stored at 2-8°C. A pharmacist or appropriately qualified designated person will be responsible for storing the APL-2 appropriately; dispensing the vials of APL-2 to the subject, study nurse, or other study personnel, and for maintaining accountability records.

## 8.3.1.3 Accountability

Records will be made of the receipt and dispensing of APL-2 for administration both on and offsite.

At the conclusion of the study, any unused investigational product will either be destroyed at the investigator site or be returned to the Sponsor or designee for destruction, and destruction will be documented appropriately. If no supplies remain, this fact will be documented appropriately.

#### 8.3.2 Planned Dose Levels and Dosing Schedule

Starting on Day 1 (Visit 3), subjects will receive SC APL-2 daily for up to 364 days.

Planned doses will be as follows:

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

| Cohort | Planned dosing schedule |
|---|---|
| Single cohort | 270 mg/day (up to 360 mg/day from Day 29) from Day 1 to Day 364* |

<sup>\*</sup> The dose may be increased up to 360 mg/day during Part 2A if the clinical response is sub-optimal. The volume to be administered will depend on the final concentration provided and will be administered as a SC infusion.

The dose for this study was determined based on safety, PK, and PD data from the ongoing studies in PNH patients.

Intra-subject dose escalations will be agreed by the Investigator and Sponsor and will be implemented on an individual subject basis and not necessarily applied across all subjects in the cohort. The dose for an individual subject will not exceed 360 mg/day (estimated to reach approximately 85 % of the  $C_{\text{max}}$  of the NOAEL observed in monkeys) without a protocol amendment.

## 8.3.3 Drug Administration

All doses will be administered as SC infusions.

The preferred site of injection will be the abdomen; however, if a subject does not tolerate administration into the abdomen alternative sites may be selected e.g. thigh or upper arm. Subjects will self-administer the SC infusions after receiving appropriate training by a research nurse or other study personnel. The injections will be administered at the clinic on those days when a clinic visit occurs and at an off-site location convenient to the subject on all other days.

Doses will be administered while subjects are seated.

Dosing records will be maintained at the clinical site and available for review by the sponsor.

#### 8.4 Concomitant Medications

#### 8.4.1 Prophylactic antibiotics

Prophylactic antibiotic therapy will be prescribed to all subjects to minimize potential infection risk. Prophylactic antibiotics will be initiated on day 1 following administration of APL-2 dosing and continue until 2 weeks after the last dose.

## 8.4.1.1 Primary prophylactic antibiotic Day 1-14

 Ciprofloxacin 500 mg twice daily, initial administration on Day 1 will take place at the initial APL-2 dosing, following ECG collection postdose.

## 8.4.1.2 Primary prophylactic antibiotic Day 15 onwards

Penicillin V 500 mg twice daily

Serious and occasionally fatal hypersensitivity (anaphylactic) reactions have been reported in patients on beta-lactam antibiotic (e.g. penicillin, amoxicillin, etc.) therapy. These reactions are more likely to occur in individuals with a history of penicillin hypersensitivity. Before initiating therapy with penicillin V, careful inquiry should be made concerning previous hypersensitivity reactions to penicillins or cephalosporins. If subjects have a known hypersensitivity to penicillin/amoxicillin they may be prescribed an alternative antibiotic at the outset.

Other frequently reported adverse effects in patients taking penicillin are diarrhea/loose stools, nausea, skin rashes and urticaria, and vomiting. Patients should, therefore, be advised that these reactions may occur.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

## 8.4.1.3 Alternative prophylactic antibiotics

- Erythromycin 500 mg twice daily
- Azithromycin 500 mg 3 times per week

Erythromycin 500 mg twice daily or Azithromycin 500 mg 3 times per week may be considered as suitable alternatives in subjects who are unable to tolerate penicillin.

The PI will discuss and agree to a suitable alternative with the sponsor's medical monitor. The agreement will be noted in the subject's medical records.

#### 8.4.2 Rescue antibiotics

Body temperature, vital signs and relevant blood parameters will be monitored regularly throughout the study to assess for signs of infection. The PI should be contacted immediately in the event of a suspected infection despite prophylactic antibiotic treatment for guidance and appropriate action to be taken. Action to be taken may include administration of a broad spectrum antibiotic to cover possible resistant organisms such as resistant pneumococcus (e.g. levofloxacin).

#### 8.4.3 Vaccinations

Vaccination against Neisseria meningitides types A, C, W, Y and B, Streptococcus pneumoniae and Haemophilus influenzae Type B (Hib) is required to participate in this study, either within 2 years prior to Day 1 dosing, or within 14 days after starting treatment with APL-2.

If required i.e. not previously vaccinated subjects will receive vaccinations against Neisseria meningitides types A, C, W, Y and B, Streptococcus pneumoniae and Haemophilus influenzae Type B (Hib). If the subject's first documented *Neisseria meningitidis* vaccine/s are administered at Day 15, a booster (for both vaccinations) should be administered after 2 months. If Pneumococcal vaccination is required, a dose of PCV13 will be administered at Day 15 and a dose of PPSV23 will be administered at least 8 weeks later (unless documented evidence exists that subjects are non-responders to vaccination as evidenced by titers or display titer levels within acceptable local limits). The PI will discuss with the Sponsor in regard to specific patient requirements

## 8.4.4 Iron Supplements

For subjects receiving iron supplements at the time of APL-2 initiation, iron supplement doses should be maintained stable throughout the study unless iron levels (ferritin and TIBC) increase to unaccepatable levels above ULN during the study. Change in dose of iron supplementation should be discussed with the Sponsor prior to implemntation

## 8.4.5 Phlebotomy/Venesection for iron overload

Phlebotomy/Venesection should only be considered if the Hb is within the normal range and may only be initiated if the need and frequency have been discussed and agreed to with the Sponsor.

## 9. STUDY PROCEDURES

Please see the Study Flow Chart in Section 2 for a summary of the schedule of study participation and procedures. The schedule of visit dates should be established, either, prior to, or at the time of screening allowing subjects an opportunity to assess whether there are likely to be significant conflicts with other activities or planned absences. To the extent possible, subjects will be expected to adhere to the visit schedule and any re-scheduling of visits must be agreed, in advance, with the investigator and sponsor to ensure that the dosing of study medication can continue daily as required.

If a subject's dose is increased beyond 270 mg/day in Part 2B additional site visits will be scheduled for the first 6 weeks of dose increase, alternating with the monthly visits in the protocol.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

i.e. subjects will return to the clinical site every two weeks for 6 weeks. These will be scheduled by the investigator and the same procedures as the monthly visits will be performed. These visits will be recorded as unscheduled visits.

## 9.1 Screening

Screening will begin within 30 days prior to dosing to confirm that subjects meet the subject selection criteria for the study. Informed consent will be obtained at screening (see Section 13.3.3). Subjects will have to meet all eligibility criteria before being enrolled into the study (see Section 7).

The following will be recorded at screening: medical history and demographic data, including, sex, age, race, body weight (kg), height (cm).

Screening procedures are listed in the Study Flow Chart in Section 2.

## 9.2 Part 1 - Treatment Period – (Days 1 to 28)

Subjects will receive daily SC doses of APL-2 on Days 1 to 28. APL-2 will be administered at the clinical site by study personnel during the first 3 days and thereafter by the subject under supervision whilst at the clinical site or off-site self-administered by the subject. Subjects will be trained to prepare and administer their infusions of APL-2, complete the administration diary and injection site assessment.

## 9.2.1 On Site Administration (Day 1 to Day 3 and Days 8, 15 and 22)

The first 3 daily SC doses of APL-2 (Day 1 to 3) will be administered by study personnel. Doses on 8, 15 and 22 will be administered, by the subject under supervision, at the clinical site. Subjects will remain in the clinic for at least 2.5 hours after receiving the first dose of APL-2 on Day 1.

If required subjects will receive vaccinations on Day 15 with boosters scheduled appropriately. Antiobiotic therapy will be changed from ciprofloxacin to penicillin V.

Blood samples for laboratory analysis, PK/PD, and antigenicity will be taken during site visits as outlined in the Study Flow Chart in Section 2.

Specific procedures for each visit are listed in the Study Flow Chart.

## 9.2.2 Outpatient Administration (Day 4 to Day 28)

From Day 4 to Day 28 daily doses of APL-2 will be self-administered by the subject at home with the exception of Days 8, 15 and 22 (see above).

Subjects will be trained to notify the PI or other study personnel in the event that an injection site reaction occurs after self-administration of APL-2. All clinically significant findings, as determined by the investigator, from injection site or related to pump use will be recorded as AEs.

## 9.3 Part 2A - Treatment Period – (Days 29 to 84)

Each subject will receive daily SC doses of APL-2 on Days 29 to 84. APL-2 will be administered by the subject. If a clinical benefit is not observed, treatment will stop on Day 28. The subject will skip Part 2A and enter Part 3 for safety follow up visits.

## 9.3.1 On Site Administration (Days 29, 36, 43, 57 and 71)

Daily SC doses of APL-2 on Days 29, 36, 43, 57 and 71 will be administered at the clinical site by the subject.

Blood samples for laboratory analysis, PK/PD and antigenicity will be taken during site visits as outlined in the Study Flow Chart in Section 2.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

Specific procedures for each visit are listed in the Study Flow Chart.

## 9.3.2 Outpatient Administration (Day 30 to Day 84)

From Day 30 to Day 84 daily doses of APL-2 will be self-administered by the subject at an off-site location convenient to the subject, with the exception of Days 36, 43, 57 and 71 (see above) where the dose will be administered at the clinical site by the subject.

## 9.4 Part 2B - Treatment Period – (Days 85 to 364)

Each subject will receive daily SC doses of APL-2 on Days 85 to 364. APL-2 will be administered at the site by the subject. If a clinical benefit is not observed, treatment will stop on Day 84. The subject will skip Part 2B and enter Part 3 for safety follow up visits.

# 9.4.1 On Site Administration (Days 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337)

Daily SC doses of APL-2 on Days 85, 113, 141, 169, 197, 225, 253, 281, 309, and 337 will be administered at the clinical site by the subject.

Blood samples for laboratory analysis, PK/PD and antigenicity will be taken during site visits as outlined in the Study Flow Chart in Section 2.

Specific procedures for each visit are listed in the Study Flow Chart.

## 9.4.2 Outpatient Administration (Day 85 to Day 364)

From Day 85 to Day 364 daily doses of APL-2 will be self-administered by the subject, with the exception of Days when the subject attends clinic visits (see above).

## 9.5 Part 3 - Follow-up - (Days 365, 379, and 393)

All subjects that complete Part 2B of the study will be asked to return to the clinical facility in Part 3 for follow-up visits on Days 365, 379, and 393. All subjects that complete Part 2A but do not enter Part 2B of the study will be asked to return to the clinical facility in Part 3 for follow-up visits on Days 85, 99 and 113. All subjects that are not eligible to enter Part 2A of the study will be asked to return to the clinical facility in Part 3 for follow-up visits on Days 29, 43 and 57.

Specific procedures including blood collection for laboratory analysis, PK/PD and antigenicity for each visit are listed in the Study Flow Chart.

## 9.5.1 Exit Visit (Day 414, or Day 134, or Day 78)

All subjects will be asked to return to the clinical facility for the Exit Visit 7 weeks after the final dose of APL-2.

Study participation for each subject will be concluded following completion of the Exit Visit. Subjects that complete Part 2B and Part 3 of the study will attend an Exit Visit on Day 414. Subjects that are not eligible to enter Part 2B but complete Part 2A of the study will attend an Exit Visit on Day 134. Subjects that are not eligible to enter Part 2A but complete Part 3 of the study will attend an Exit Visit on Day 78. If a subject withdraws from the study prior to the scheduled Exit Visit, all Exit Visit evaluations should be performed at the subject's final visit to the clinic, including the collection of blood samples for PK and/or PD assessments, as well as a post-dose antigenicity sample if not yet collected.

The Exit Visit procedures are listed in the Study Flow Chart in Section 2.

## 9.5.2 Unscheduled Follow-up Visits

All subjects will be asked to return to the clinical facility for additional follow-up visits if considered necessary by the PI or if PK/PD sampling schedule is modified or extended based on interim results.

Unscheduled follow-up visits may include any of the procedures listed in the Study Flow Chart in Section 2.

## 9.5.3 Scheduled End of Study

The end of the study is scheduled after completion of the Exit Visit evaluations.

## 9.6 Periodic Safety Review

A periodic safety review will take place on a regular (approximately bi-monthly) basis as detailed below.

## 9.6.1 Safety Monitoring Committee

A Safety Monitoring Committee (SMC) will review cumulative safety/tolerability data (e.g., physical examinations, ECGs, vital signs, clinical laboratory tests, and adverse events [AEs]), efficacy (LD levels, haptoglobin levels, Hb levels, reticulocyte counts, and RBC transfusions) and PK data including predicted exposures based on emerging PK data. The SMC will have the responsibility to conduct a thorough safety assessment at regular intervals during the treatment phase of the study. A key responsibility of the SMC will be to decide whether to continue or modify the study based on recommendations by the sponsor and upon an evaluation of emerging safety and efficacy data. The first SMC meeting will be scheduled within 3 months after the first subject is randomized, and a future intervals presented within the SMC charter. Regular or *ad hoc* SMC data reviews may be recommended by the SMC or requested by the Sponsor.

If efficacious and safe, APL-2 may reduce LD levels, improve Hb levels and reduce transfusion dependency in these patients. The SMC will be responsible for reviewing individual subject data to understand if there is a health benefit in these individuals at any time during the treatment period. If a benefit is observed the SMC may recommend extending the treatment beyond 364 days either through a protocol amendment or an extension study.

The remit, roles, and responsibilities of the SMC will be specified in a separate SMC charter.

## 9.7 Removal of Subjects from the Study

Subject participation in this study may be discontinued for any of the following reasons:

- Occurrence of any medical condition or circumstance that exposes the subject to substantial risk and/or does not allow the subject to adhere to the requirements of the protocol.
- 2. Any SAE, clinically significant AE, severe laboratory abnormality, intercurrent illness, or other medical condition that indicates to the PI that continued participation is not in the best interest of the subject.
- 3. Subject's decision to withdraw.
- 4. Subject failure to comply with protocol requirements or study-related procedures.
- 5. Termination of the study by the Sponsor, FDA, or other regulatory authorities.

The clinical report will include reason(s) for subject withdrawals as well as details relevant to the subject withdrawal. If a subject is withdrawn from the study prior to study completion, the subject will undergo all procedures scheduled for study completion (Exit Visit) as the situation allows. Any

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 
subject withdrawn due to an AE (whether serious or non-serious) or clinically significant abnormal laboratory test values will be evaluated by the PI or a monitoring physician and will be treated and/or followed up until the symptoms or values return to normal or acceptable levels, as judged by the PI.

Subjects who are withdrawn may be replaced. Replacement of subjects will be discussed on a case by case basis.

#### 10. ASSESSMENTS

#### 10.1 Assessments

Assessments to be performed during the study are described below. Every effort should be made to ensure that the protocol-required assessments are completed as described.

If deemed necessary, additional safety measurements will be performed at the discretion of the PI.

## 10.1.1 Body Height and Weight

Body height (cm) and body weight (kg) will be measured at screening as part of the physical examination.

#### 10.1.2 Physical Examination

All physical examinations will include, at a minimum, assessment of the following: general, head, ears, eyes, nose and throat, dentition, thyroid (endocrine), heart, chest, lungs, abdomen, skin, extremities, back/neck, musculoskeletal, and lymph nodes.

A licensed physician employed at the study site will examine each subject as outlined in the Study Flow Chart in Section 2.

Medical history will be recorded at screening.

A symptom-driven physical examination may be performed at various unscheduled time points if deemed necessary by the PI.

#### 10.1.3 Vital Signs

Single measurements of body temperature, respiratory rate, blood pressure, and heart rate will be measured as outlined in the Study Flow Chart in Section 2.

Vital signs may be taken at any other times, if deemed necessary. Blood pressure and heart rate measurements will be performed with subjects in a seated position after resting for 5 minutes, except when they are supine or semi-reclined because of study procedures and/or AEs (e.g., nausea, dizziness) or if deemed necessary by the PI.

Vital signs will be measured before venipuncture and ECG.

At clinic visits vital signs will be measured pre- and post-dose. Vital signs will be measured within 2 hours prior to dosing for the pre-dose time point. Post-dose vital signs readings will be performed within approximately 30 minutes after dosing.

## 10.1.4 Electrocardiogram Monitoring

Single 12-lead ECGs will be done at the time points outlined in the Study Flow Chart in Section 2.

If done on dosing days, ECGs will be performed within approximately 30 min after dosing.

ECGs will be taken following resting in the supine position for 10 min in a guiet environment.

ECGs will be interpreted and signed and dated by the PI. The ECGs will be classified as normal, having a not clinically significant (NCS) abnormality, or having a clinically significant (CS)

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

abnormality. In addition, ECG parameters of ventricular rate, PQ or PR interval, QRS duration, and QT interval (corrected using both Bazett's and Fridericia's method and uncorrected) will be noted on the CRF. All CS findings will be recorded as AEs.

# 10.1.5 Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale

The FACIT Fatigue Scale is a 13 item Likert scaled instrument which is self-administered by the subjects during clinic visits on as outlined in the Study Flow Chart in Section 2. The subject is presented with 13 statements and is asked to indicate their response as it applies to the past 7 days. The 5 possible responses are 'Not at all' (0), 'A little bit (1), 'Somewhat' (2), 'Quite a bit' (3) and 'Very much' (4). With 13 statements the total score has a range of 0 to 52. Before calculating the total score, some responses are reversed to ensure that the higher score corresponds to a higher quality of life. The FACIT Fatigue Scale and scoring guidelines are provided in the Manual of Procedures (MOP).

## 10.1.6 Linear Analog Scale Assessment (LASA) for Quality of Life

The Linear Analog Scale Assessment (LASA) consists of three items asking respondents to rate their perceived level of functioning. Specific domains include activity level, ability to carry out daily activities, and an item for overall QOL. A representation of the scale is presented in Appendix 2 (see Appendix 2). LASA is self-administered by the subjects during clinic visits as outlined in the Schedule of Events in Section 2. Scores for the three individual components of the scale and the combined score will be included in the analysis and this will be described in the Statistical Analysis Plan.

#### 10.1.7 Clinical Laboratory Tests

All tests listed below will be performed as outlined in the Study Flow Chart in Section 2. In addition, laboratory safety tests may be performed at various unscheduled time points, if deemed necessary by the PI or recommended by the SMC. The clinical laboratory tests include (but are not limited) the following:

#### **10.1.7.1 Hematology**

- Hb
- Hematocrit
- RBC count

## 10.1.7.2 Coagulation

- Prothrombin time (PT)
- Fibrinogen

## 10.1.7.3 Serum Chemistry

- Blood urea nitrogen (BUN)
- Creatinine
- Estimated creatinine clearance (using Cockcroft-Gault formula) – screening only
- Bilirubin (total and direct)
- Albumin

- Platelet count
- WBC count with differential
- Reticulocytes
- Activated partial thromboplastin time (aPTT)
- D-Dimer
- Aspartate aminotransferase (AST)
- ALT
- Uric acid
- Glucose
- Sodium

- Alkaline phosphatase (ALP)
- Lactate dehydrogenase (LD)
- Haptoglobin
- Gamma-glutamyl transpeptidase (GGT)
- Creatine kinase (CK)

- Potassium
- Chloride
- Ferritin
- B12/folate
- Total Iron Binding Capacity (TIBC)

## 10.1.7.4 Urinalysis

- pH
- Specific gravity
- Protein
- Glucose
- Ketones

- Bilirubin
- Blood
- Nitrite
- Urobilinogen
- Leukocyte esterase

If an abnormality is noted for protein, blood, nitrite and/or leukocyte esterase, a microscopic examination will be performed.

## 10.1.7.5 Human Chorionic Gonadotropin (Serum Pregnancy Test) and Follicle-Stimulating Hormone

Serum Pregnancy Test will be performed for females only. FSH will be performed for postmenopausal females at screening only.

## 10.1.8 Injection/ Infusion Site and Pump Safety Assessment

On the days of clinical visits, an assessment of the APL-2 injection site, and pump use safety will be performed within 30 minutes after study drug administration. The assessment will be performed by a physician or other licensed health care provider (e.g. study nurse) as delegated by the investigator. The injection site and the surrounding area will be inspected for redness, swelling, induration, and bruising; and the subject will be asked about the presence of pain and/or tenderness, and any issue related to pump use. The date, time, and outcome of the injection site assessment will be recorded on the source documents and CRFs.

Subjects will be trained to notify the PI or other study personnel in the event that an injection site reaction occurs after self-administration of APL-2. All clinically signficant findings, as determined by the investigator, from injection site or related to pump use will be recorded as AEs.

#### 10.2 Pharmacokinetic Assessments

#### 10.2.1 Blood Sampling and Processing

Blood samples for PK assessment of APL-2 will be collected via direct venipuncture at the time points delineated in the Study Flow Chart in Section 2.

On Day 1 only, a PK sample will be taken pre-dose and at a minimum of 2.5 hours post-dose (or later depending on how long the subject is kept at the clinic). All PK samples on other study days will be collected pre-dose.

Instructions for collection, handling, processing, storage, and shipping of samples will be provided in a separate sample handling manual prior to study initiation.

#### 10.2.2 Analytical Method

Serum sample analysis will be performed using GLP-compliant validated procedures and methods. The methods used and the results obtained will be included in the final report as an appendix.

## 10.3 Flow Cytometry Assessments

Blood samples will be collected via direct venipuncture at the time points delineated in the Study Flow Chart in Section 2. Flow cytometry assessment will include, but not be limited to: PNH clonal distribution of RBCs, CD71+ immature reticulocytes, monocytes and granulocytes and C3 deposition on RBCs.

Instructions for collection, handling, processing, storage, and shipping of samples will be provided in a separate sample handling manual prior to study initiation.

#### 10.4 Pharmacodynamic Assessments

Blood samples will be collected via direct venipuncture at the time points delineated in the Study Flow Chart in Section 2. for PD assessment of complement activation through the classical (e.g., CH50) and alternative (e.g., AP50) pathways. Blood samples will also be collected to measure C3 levels. Other relevant PD markers may also be assessed.

Instructions for collection, handling, processing, storage, and shipping of samples will be provided in a separate Laboratory Reference Manual prior to study initiation.

#### 10.5 Anti- APL-2 Antibody Assessment

Patients who test positive for anti-APL-2 antibodies at any time will be followed with ADA samples being collected every 6 months until the antibody levels revert to baseline. Samples that test positive will be characterized by an assay that will determine antibody titer, binding to the cyclic peptide or PEG domains, and measure neutralizing capacity.

The proposed ADA sampling schedule was established to capture the ADA signal at baseline, along with any potential early onset and the dynamic profile (transient or persistent) of antibody formation while minimizing APL-2 level in the sample.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

#### 10.6 Blood Volume for Study Assessments

Table 2: Blood Volume during Study (up to Day 414)

| Assay | Number of<br>Time Points | Approximate<br>Volume per<br>Time Point *<br>(mL) | Approximate Sample<br>Volume Over Course<br>of Study (mL) |
|---|---|---|---|
| Pharmacokinetics | 19 | 2 | 38 |
| Anti-APL-2 Ab assay | 9 | 2 | 18 |
| Hematology | 20 | 3 | 60 |
| Chemistry (Incl. screen serology and pregnancy) | 20 | 3 | 60 |
| Coagulation profile | 20 | 4.5 | 90 |
| Complement profile (C3, CH50 and AP50) | 20 | 4 | 80 |
| Flow cytometry for PNH and C3 deposition | 20 | 2 | 40 |
| Plasma Hb | 20 | 4 | 80 |
| Total Approximate Blood Volui | 466** | | |

 <sup>\*</sup> Represents the largest collection volume planned over the duration of the study (smaller tubes will be used whenever possible).

## 10.7 Pregnancy tests

For WOCBP, a serum pregnancy test will be performed at screening, and subjects with a positive test will be excluded from the study. A follow up urine pregnancy test will be performed on Day 1 pre-dose (a negative urine pregnancy test must be received before dosing with study drug). A urine pregnancy test will also be performed at each site visit (pre-dose) if applicable. A final urine pregnancy test will be performed at the final Exit Visit. Male subjects will be counseled to avoid donating sperm after dosing on Day 1 until the final Exit Visit.

#### 11. ADVERSE EVENTS

#### 11.1 Definitions

An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign, including a clinically significant abnormal laboratory finding, symptom, or disease temporally associated with the use of a study drug, whether or not considered related to the study drug.

Adverse events include the onset of new illness and the exacerbation of pre-existing conditions. Any medical condition that is present at the time that the subject is screened should be recorded on the medical history eCRF and not reported as an AE. However, if that condition deteriorates or severity changes at any time during the study, it should be recorded as an AE.

Any AEs that occur prior to dosing on Day 1 will be categorized as pre-treatment events. Treatment-emergent adverse events (TEAEs) will be defined as those AEs that occur after dosing on Day 1 and up to 30 days after the last dose of study medication.

A suspected adverse reaction means any AE for which there is a reasonable possibility that the drug caused the AE. Reasonable possibility means there is evidence to suggest a causal relationship between the drug and the AE.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

<sup>• \*\*</sup> If dose is increased to 360 mg/day, additional blood draws will be scheduled.

#### 11.2 Recording Adverse Events

Subjects will be monitored for adverse events throughout the study. Adverse events may be volunteered spontaneously by the study subject, or discovered by the study staff during physical examinations, or by asking open, non-leading questions (e.g. "How have you been feeling since the last clinic visit?"). Subjects will be instructed to inform the investigator and/or study staff of any AEs that may occur at any time during the study.

All AEs occurring from screening through the final Exit visit will be recorded in detail in the source documents and documented on the appropriate AE or SAE eCRF. The nature of the AE, date (and time, if known) of AE onset, duration, severity, and action taken will be documented, together with the Pl's assessment of the seriousness of the AE and relationship to study drug. All AEs should be recorded in the study subject's own words (verbatim), unless in the opinion of the PI, the AE constitutes a recognized condition, disease, or syndrome. In that case, the condition, disease or syndrome should be named rather than the individual symptoms. The AEs will be coded using the current Medical Dictionary for Regulatory Activities (MedDRA).

Outcome will be recorded as:

- Ongoing
- Resolved
- · Resolved with sequela
- Death or
- Unknown

#### 11.3 Assessment of Adverse Events

Each AE will be assessed by the PI or physician designee with regard to the categories discussed in the sections below.

#### 11.3.1 Intensity

The PI will determine the severity of each AE. AEs will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. The following definitions for rating severity will be used:

| Grade 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. |
|---|---|
| Grade 2 | Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL)*. |
| Grade 3 | Severe or medically significant but not immediately life-<br>threatening; hospitalization or prolongation of hospitalization<br>indicated; disabling; limiting self-care ADL**. |
| | Note: An experience may be severe but may not be serious, e.g., severe headache). |
| Grade 4 | Life-threatening consequences; urgent intervention indicated. |
| Grade 5 | Death related to AE |

- A semi-colon indicates 'or' within the description of the grade.
- \*Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.
- \*\*Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

When changes in intensity of an AE occur more frequently than once a day, the maximum intensity for the event should be noted for that day. Any change in severity of signs and/or symptoms over a number of days will be captured and recorded as a new AE, with the amended severity grade, and the date and time (if known) of the change.

## 11.3.2 Causality

The relationship of an AE to the study drug will be assessed using the following criteria:

| Definitely<br>Related | <ul> <li>Event or laboratory test abnormality, with plausible time relationship to drug intake</li> <li>Cannot be explained by disease or other drugs</li> <li>Response to withdrawal plausible (pharmacologically, pathologically)</li> <li>Event definitive pharmacologically or phenomenologically (i.e. an objective and specific medical disorder or a recognized pharmacological phenomenon)</li> <li>Rechallenge satisfactory, if necessary</li> </ul> |
|---|---|
| Possibly<br>Related | <ul> <li>Event or laboratory test abnormality, with reasonable time relationship to drug intake</li> <li>Could also be explained by disease or other drugs</li> <li>Information on drug withdrawal may be lacking or unclear</li> </ul> |
| Unlikely<br>Related | <ul> <li>Event or laboratory test abnormality, with a time to drug intake that makes a relationship improbable (but not impossible)</li> <li>Disease or other drugs provide plausible explanations</li> </ul> |
| Not Related | <ul> <li>Event or laboratory test abnormality, is plausibly related to the participant's clinical state, underlying disease, or the study procedure/conditions</li> <li>Time relationship to drug intake makes a relationship unreasonable</li> <li>Other obvious causes for event or laboratory test abnormality exist</li> </ul> |
| Unknown | <ul> <li>Report suggests an adverse event, however, cannot be judged at this time because information is insufficient or contradictory</li> <li>More data for proper assessment is needed, or additional data is under examination</li> </ul> |

#### 11.3.3 Serious Adverse Event

A serious adverse event (SAE) is defined as any untoward medical occurrence that at any dose:

- Results in death;
- Is life-threatening: this means that the subject was at risk of death at the time of the event; it
  does not mean that the event might have caused death had it occurred in a more severe
  form:
- Required hospitalization or prolongation of existing hospitalization;
- Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions;
- Is a congenital anomaly or birth defect.

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in the above definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

Medical and scientific judgment should be exercised in deciding if an AE is serious and if expedited reporting is appropriate.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

#### 11.4 Reporting Serious Adverse Event

The reporting period for adverse events begins as soon as the subject's written consent to participate in the study has been obtained, and continues through the final Exit visit, or 30 days after the final dose of study medication. The PI is responsible for reporting all SAEs to the Safety Monitor, whether or not the event is considered related to the study drug.

If an SAE occurs, the PI should complete and sign the SAE Report Form, and fax or email it to the Safety Monitor at the number/address which will be provided separately to the investigator sites, within 24 hours of becoming aware of the event:

The initial SAE Report should include, at a minimum, the following information:

- Study number
- Subject number/ID
- Gender
- Date of birth
- Name of PI and full clinical site address
- Details of SAE
- Criterion for classification as "serious"
- Study drug name and treatment start date
- Date of SAE onset
- Causality assessment (if sufficient information is available to make this determination)

The Safety Monitor, or designee, will request clarification of omitted or discrepant information from the initial report. The PI or designee is responsible for emailing or faxing the requested information to the Safety Monitor within 24 hours of the request.

Initial reports of SAEs must be followed later with detailed descriptions, including clear copies of supporting documents as necessary (e.g. hospital discharge summary, laboratory reports, autopsy reports, etc.), with the subject's personal identifiers removed. If a new SAE Report Form is faxed, the PI must sign and date the form.

The PI must report all SAEs to the IRB/IEC according to the institutional IRB/IEC policy.

## 11.5 Adverse Events of Special Interest

An adverse event of special interest is one of scientific and medical concern specific to the Sponsor's product or program where ongoing monitoring and rapid communication by the PI to the Sponsor may be appropriate. These adverse events may be serious or non-serious. Applicable adverse events may require further investigation in order to characterize and understand, and depending upon the nature of the event, rapid communication by the trial Sponsor to other parties may also be required. These adverse events of special interest must be reported promptly to the sponsor. The adverse events of special interest include the following:

- Local or systemic infection of any origin
- Thrombosis
- Clinically significant decrease in kidney function
- Injection site reactions

If an adverse event of special interest occurs in a study subject, the study subject will be followed for resolution of the adverse event. A decision will be made by the Sponsor concerning further exposure to the study treatment and further participation in the study.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

## 11.6 Unexpected Adverse Events or Unexpected Suspected Adverse Reactions

An AE or suspected adverse reaction is considered "unexpected" if it is not listed in the Investigator's Brochure (IB) or is not listed at the specificity or severity that has been observed; or is not consistent with the risk information described in the general investigational plan or elsewhere in the current application. For example, under this definition, hepatic necrosis would be unexpected (by virtue of increased severity) if the IB referred only to elevated hepatic enzymes or hepatitis.

The Sponsor will be responsible for reporting any serious and unexpected adverse events to the applicable regulatory agencies as required.

## 11.7 Treatment and Follow up of Adverse Events

AEs (whether serious or non-serious), including clinically significant abnormal laboratory test values, will be evaluated by the Investigator and treated and/or followed up until the symptoms or value(s) return to baseline or are clinically stable. Treatment of AEs will be performed by appropriately trained medical personnel, either at the clinical site or at a nearby hospital emergency room. When appropriate, medical tests and/or examinations will be performed to document resolution of the event(s).

AEs continuing after completion of the study will be followed up by telephone or with visits per the discretion of the PI. If possible, the outcome of any AE that caused discontinuation from the study or was present at the end of the study should be reported, particularly if the AE was considered by the PI to be related to the study drug.

## 11.8 Pregnancy

Although pregnancy is not considered an AE, the outcome of a pregnancy, if there is a spontaneous abortion, congenital anomaly or other adverse fetal outcome, may be an SAE. All SAEs are to be reported to the study sponsor on the SAE Reporting Form. Pregnancies will be reported using a pregnancy report form.

WOCBP and males with female partners of child-bearing potential will be instructed to practice an acceptable method of birth control (as defined in Section 7.1.1) for the duration of the study.

If a female subject or partner of a male subject becomes pregnant during the study, the PI should report the pregnancy to the Safety Monitor within 24 hours of being notified. The subject or partner should be followed by the PI until completion of the pregnancy. At the completion of the pregnancy, the PI will document and report the outcome. If the outcome of the pregnancy meets the criteria for classification as an SAE (i.e. postpartum complication, stillbirth, neonatal death, or congenital anomaly) the PI should follow the procedures for reporting an SAE (Section 11.4).

#### 12. STATISTICS

## 12.1 Sample Size Justification

The study will be conducted alongside the ongoing Phase Ib study APL2-CP-PNH-204 (PADDOCK) to investigate APL-2 in PNH patients who have not previously received treatment with eculizumab. Safety and efficacy data from both studies will be used to support the data obtained in the Phase III confirmatory study. Up to 20 subjects will be enrolled to complete 28 days of dosing. The sample size is considered sufficient to obtain useful safety, tolerability, PD and PK data to support the clinical program.

#### 12.2 Statistical Analysis Methodology

A formal Statistical Analysis Plan (SAP) will be developed and finalized prior to locking the database. The full details of data presentations and analyses will be provided therein. Additional statistical analyses other than those described in this section may be performed if deemed

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

appropriate and included in the SAP. Any deviations from the final analysis plan or from what is outlined in the protocol will be discussed in the final study report.

No formal inferential statistics will be applied to data collected in the study.

The data from this study will also be pooled with the Cohort 2 data from the Phase Ib study APL2-CP-PNH-204 (PADDOCK), which also investigates 270mg/day APL-2 in PNH patients who have not previously received treatment with eculizumab. The details of reporting this pooled data will be documented in a separate SAP.

#### 12.2.1 Analysis Populations

#### 12.2.1.1 Screened Population

The Screened Population will include all subjects who signed the informed consent form and are screened for participation in this study. This set will be used only for the purpose of describing subject disposition.

## 12.2.1.2 Safety Population/ Intent to Treat (ITT) Population

The Safety Population will include all subjects eligible to receive study medication and who receive at least one dose of study medication. The Intent to Treat Population will be identical to the Safety Population for this study. All baseline characteristics, demographic and efficacy endpoint data will be presented using the ITT Population.

#### 12.2.1.3 Pharmacokinetic (PK) Population

The PK Population will include all subjects in the Safety Population who have at least one quantifiable concentration of APL-2.

#### 12.2.1.4 Pharmacodynamic (PD) Population

The PD Population will include all subjects in the Safety Population who have at least one quantifiable post dose PD parameter.

#### 12.2.1.5 Data Review for Analysis Populations

After all the data have been verified/coded/entered into the database, a review will be performed. The purpose of this review will be to define the analysis populations. The review will also check the quality of the data, identifying outliers, and making decisions on how to deal with problems in any data (e.g., missing values, withdrawals, protocol deviations). After the pre-analysis review, resolution of all issues and documentation of all decisions, the database will be locked.

#### 12.2.2 Study Endpoints

#### 12.2.2.1 Safety Endpoints

The primary safety endpoints of the study are the number and severity of TEAEs. Safety will also be assessed through vital signs, 12-lead ECG and laboratory safety data. Changes from baseline will be calculated using the last measurement prior to the start of dosing as baseline.

#### 12.2.2.2 Efficacy Endpoints

Changes from baseline and percentage changes from baseline in LD, haptoglobin and Hb are the primary efficacy endpoints. They will be calculated for each post dose assessment, where the baseline will be taken as the last measurement prior to the start of dosing.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

#### 12.2.2.3 Secondary Endpoints

Secondary endpoints include:

- changes from baseline in FACIT Fatigue Scale (Version 4)
- · changes from baseline and percentage changes from baseline in reticulocyte count
- changes from baseline and percentage changes from baseline in total bilirubin
- changes from baseline in the number of RBC transfusions per month and number of units transfused per month
- changes from baseline in LASA scale scores (individual and combined).

Baseline will be taken as the last measurement prior to the start of dosing. For transfusions baseline will be taken from the 12 month transfusion history.

## 12.2.2.4 Pharmacokinetic Endpoints

Plasma concentrations of APL-2 will be determined from multiple samples taken between Day 1 and the Exit Visit.

## 12.2.2.5 Exploratory Pharmacodynamic Endpoints (Markers)

Changes from baseline and percentage changes from baseline will be calculated for each of the complement parameters (CH50, AP50 and C3), C3 deposition on RBC cells and clonal distribution of PNH RBCs. Baseline will be taken as the last measurement prior to the start of dosing.

#### 12.2.3 Safety Analyses

All safety endpoints will be evaluated using the Safety Population.

#### 12.2.3.1 Adverse Events

Treatment emergent adverse events (TEAE) are defined as those AEs that develop or worsen after the first dose of study medication and up to 30 days beyond the last dose of study medication. The current version of Medical Dictionary for Regulatory Activities (MedDRA) will be used to classify all AEs.

TEAE will be summarized by system organ class and preferred term. Tabulations will be produced for all TEAEs, for those considered potentially treatment related (causality to study drug is reported as possibly or probably, or where causality is not reported) and for TEAE of special interest. Number of subjects reporting SAEs will also be tabulated.

A by-subject TEAE data listing, including verbatim term, preferred term, treatment, severity, and investigator judgment of relationship to treatment, will be provided.

#### 12.2.3.2 Clinical Laboratory Tests

A by-subject listing will be provided including changes from baseline. Laboratory values that are outside the laboratory reference range will be flagged.

#### 12.2.3.3 Vital Signs and ECGs

Observed and change from baseline values for vital sign and ECG parameter will be listed.

Values of potential clinical significance (e.g. change in QTcF ≥30ms from baseline) will be flagged in listings and summarized.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

#### 12.2.4 Efficacy and Secondary Endpoint Analyses

The efficacy and secondary endpoints will be evaluated for the ITT Population.

Absolute values, changes from baseline and percentage changes from baseline (where appropriate) will be summarised, using descriptive statistics, by study visit. Data will be plotted by study day.

The number of RBC transfusions per month and number of units transfused per month will be summarized over the study.

## 12.2.5 Pharmacokinetic Analyses

The PK concentrations will be evaluated using the PK Population.

Individual concentration over time profile plots will be presented. Median profiles of the concentration-time data, using nominal sampling times, will also be presented. Both linear-linear and linear-log plots will be presented. APL-2 concentrations will be summarized by study visit using descriptive statistics.

Where appropriate, steady-state PK parameters for APL-2 will be estimated from the individual serum concentrations-time data, using actual sample times using a non-compartmental approach. PK parameters will include:

AUCtotal: The area under the serum concentration versus time curve, from time 0 (pre-dose Day 1) to the last measurable concentration (t) at the end of study.

Ctrough, max: Maximum observed pre-dose serum concentration.

PK parameters will be summarized using descriptive statistics.

PK data will be combined with the prior data collected in earlier clinical studies and then used to update the APL-2 population PK model (Apellis Data on File).

#### 12.2.6 Pharmacodynamic Analyses

The PD parameters will be evaluated using the PD Population.

Absolute values, changes from baseline and percentage changes from baseline will be summarised, using descriptive statistics, by study visit. Individual parameter over time profile plots will be presented. Median profiles over time, using nominal sampling times, will also be presented.

#### 12.2.7 Handling of Dropouts and/or Missing Data

No imputation of missing data for early terminations will be performed.

Where appropriate screen values may be used as baseline in the event of missing Day 1 measurements.

Missing dates/times will be reviewed on a case by case basis for potential imputations, but the original data will always be presented in data listings.

PK concentration values below the limit of quantification will take the value of 0 in individual linear-linear profile plots and the limit of quantification in linear-log profile plots.

#### 12.2.8 Other Data Analyses

Demographic data, baseline characteristics, physical examination, concomitant medication and medical history data will be listed. The current versions of the World Health Organization (WHO) and MedDRA coding dictionaries will be used for the concomitant medications and medical histories respectively.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

## 12.3 Interim Analyses

As mentioned in Section 9.6, a periodic safety review will take place on a regular basis by the SMC to review safety/tolerability, PK and PD data.

Data may be reported while the study is ongoing to help guide decisions to further develop APL-2. These reports will be performed on data that will have been fully checked and considered as final. Any changes to the data previously reported will be fully auditable and discussed in subsequent reports.

#### 13. ADMINISTRATIVE CONSIDERATIONS

#### 13.1 Direct Access to Source Data/Documents

The PI must maintain, at all times, the primary records (i.e. source documents) of each subject's data for data verification. Examples of source documents are medical records, laboratory reports, study drug records, and eCRFs that are used as the source.

The PI will permit trial-related monitoring, audits, and inspections by the Sponsor and/or its' designee, IRB/IEC, and the regulatory agencies at any time during the study. The PI will ensure that the auditor is allowed direct access to the source data, medical records, eCRFs, and the Site's regulatory file for the study and any other pertinent information.

## 13.2 Quality Control and Quality Assurance

This study is to be performed in full compliance with the protocol, Good Clinical Practices (GCP), and applicable regulatory requirements. The PI, Sponsor and/or its' designee are responsible for ensuring that the study staff receive appropriate training on the protocol, study procedures and any other relevant information.

Quality assurance and quality control systems are implemented and maintained using written Investigative site, Sponsor and/or designee Standard Operating Procedures (SOPs) to ensure that the study is conducted and data are generated, documented (recorded), and reported in compliance with the protocol, GCP, and the applicable regulatory requirement(s) and local laws, rules, regulations.

Quality control (QC) checks will be applied at each stage of data handling (e.g. edit checks) to ensure that all data are reliable and have been processed correctly.

#### 13.2.1 Monitoring

On-site monitoring will be performed by the Sponsor's designee for the duration of the study. The monitor will ensure that the study is conducted, recorded and reported in accordance with the protocol, SOPs, GCP, and the applicable regulatory requirements. The monitor will verify the accuracy and completeness of the eCRF entries, source documents, and other study-related records against each other. The PI will provide direct access to source data/documents for study-related monitoring. It is important that the PI and the staff are available at these visits. The monitor will record the date of each visit together with a summary of the status and progress of the study. Proposed actions will be documented in writing to the PI.

#### 13.3 Ethics

## 13.3.1 Ethical Conduct of the Study

This research will be carried out in accordance with the protocol, applicable regulations, the ethical princliples set forth in the Declaration of Helsinki, and the ICH Harmonized Tripartite Guidance for Good Clinical Practice, E6, R1 (ICH GCP).

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

#### 13.3.2 Institutional Review Board/Ethic Committee

The study protocol, any amendments to the protocol, informed consent form, the Investigator's Brochure, and other study specific information will be reviewed and approved by the IRB/IEC. The study will not be initiated until the IRB/IEC has approved the protocol or a modification thereof. All records pertaining to IRB/IEC submission and approval should be kept in the site's regulatory files and Sponsor's Trial Master File (TMF).

The IRB/IEC must be constituted and operate in accordance with the principles and requirements described in ICH Guidance E6 and local regulations as deemed appropriate.

#### 13.3.3 Subject Information and Consent

The PI is responsible for obtaining an informed consent. A written informed consent, in compliance with ICH Guidance E6, must be obtained from each subject prior to screening and enrollment or performing any study related procedures.

The purpose of the study, the procedures to be carried out and the potential hazards will be described to the subjects in non-technical terms. The subject will be given sufficient time to consider the study's implications before deciding to participate in the study. The subject and/or legal guardian (if permitted by local national legislation) will be required to sign and date an Informed Consent Form (ICF) and will be assured that they may withdraw from the study at any time without jeopardizing their medical care. The PI shall retain the original, signed informed consent for study participation in the subject's medical record and shall provide the subject and/or legal guardian with a copy of the signed consent.

If there are any changes/amendments to the approved protocol, which may directly affect the subject's decision to continue participation in the study, the ICF shall be amended to incorporate the changes to the protocol and the subject must re-sign the IRB/IEC approved amended ICF.

#### 13.3.4 Confidentiality

Confidentiality of subject's information must be maintained in accordance with local privacy laws.

#### 13.3.5 ClinicalTrials.gov

This study has been listed with ClinicalTrials.gov, as required.

#### 13.3.6 Termination of Study

The Sponsor reserves the right to suspend or discontinue this study for administrative and/or safety reasons at any time. The PI reserves the right to discontinue dosing subjects at any time for safety reasons.

#### 13.4 Data Handling and Record Keeping

The PI must maintain all documentation related to this study. All essential documents (as defined in the ICH Guideline E6) and the data generated in connection with this study, together with the original copy of the final report, will be retained for at least 5 years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or at least 5 years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents should be retained for a longer period if required by the applicable regulatory requirements or by an agreement with the Sponsor.

It is the responsibility of the Sponsor to inform the PI/Institution as to when these documents no longer need to be retained.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

## 13.5 Protocol Amendments

Any amendments to the study protocol deemed necessary as the study progresses will be discussed between Sponsor and the PI. The PI will not implement any changes to the protocol without an agreement by the Sponsor and prior review and documented approval from the IRB/IEC of an amendment, except where necessary to eliminate immediate hazards to study subject or when the changes involve only logistical or administrative aspects of the study (e.g., change in staff, telephone numbers).

Changes resulting in amendments will be made jointly between the Sponsor and the PI and must be confirmed in writing. Amendment(s) will be approved and signed off in the same way as the protocol.

## 13.6 Report Format

According to the ICH Harmonized Tripartite Guideline (Organization of the Common Technical Document for the Registration of Pharmaceuticals for Human Use M4 and the ICH M2 Expert Working Group), the final report will be written according to the ICH E3 Guideline (Structure and Content of Clinical Study Reports).

#### 13.7 Finance and Insurance

Finance and insurance will be addressed in a Clinical Trial Agreement between the PI/Institution and the Sponsor (or CRO authorized to enter into Clinical Trial Agreements for and on behalf of the Sponsor).

#### 13.8 Publication Policy

The data generated for this study are considered confidential information and are the property of the Sponsor. All study information provided to the PI and Site personnel by the Sponsor shall not be published or disclosed to a third party without the prior written consent of the Sponsor.

After the completion of the study, the data may be reported at a scientific meeting and/or submitted for publication in a scientific journal with the prior written consent of the Sponsor. The Sponsor must be given at a minimum 30 days to review the materials to be presented at a scientific meeting and/or for publication in a scientific journal.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

#### 14. REFERENCES

- 1. DeZern AE, Dorr D, and Brodsky, RA. Predictors of Hemoglobin Response to Eculizumab Therapy in Paroxysmal Nocturnal Hemoglobinuria, *Eur J Haematol.*, 2013, 90(1), p.16-24
- 2. Apellis Pharmaceuticals, Inc. Product: APL-2 Injection. Investigator's Brochure. Final Version 1.0. 12 June 2014.
- 3. FDA Guidance for Industry: Estimating the Maximum Safe Starting Dose in Initial Clinical Trials for Therapeutics in Adult Healthy Volunteers. July 2005. Available online: http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidance s/ucm078932.pdf
- 4. FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. September 2007. Available online:
  - http://www.fda.gov/downloads/BiologicsBloodVaccines/GuidanceComplianceRegulatoryInformation/Guidances/Vaccines/ucm091977.pdf
- 5. FDA Guidance for Industry and Investigators: Safety Reporting Requirements for INDs and BA/BE Studies-Small Entity Compliance Guide. December 2012. Available online: http://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidance s/UCM332846.pdf
- 6. Ivens, I. A., Baumann, A., McDonald, T. A., Humphries, T. J., Michaels, L. A., and Mathew, P. (2013). PEGylated therapeutic proteins for haemophilia treatment: a review for haemophilia caregivers. Haemophilia 19: 11-20
- 7. Rudmann, D.G., Alston, J.T., Hanson, J.C., and Heidel, S. (2013). High molecular weight polyethylene glycol cellular distribution and PEG-associated cytoplasmic vacuolation is molecular weight dependent and does not require conjugation to proteins. Toxicol Pathol 41: 970-983.
- 8. Walpole, S.C., Prieto-Merino, D., Edwards, P., Cleland, J., Stevens, G., and Roberts, I. (2012). The weight of nations: an estimation of adult human biomass. BMC Public Health 12 (1): 439.
- 9. GBD 2013 Mortality and Causes of Death Collaborators (2015). Global, regional, and national age—sex specific all-cause and cause-specific mortality for 240 causes of death, 1990–2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015;385(9963): 117–171.

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

# 15. APPENDIX 1: FUNCTIONAL ASSESSMENT OF CHRONIC ILLNESS THERAPY (FACIT) FATIGUE SCALE

## **FACIT Fatigue Scale (Version 4)**

Below is a list of statements that other people with your illness have said are important. Please circle or mark one number per line to indicate your response as it applies to the <u>past 7 days</u>.

| | | Not at<br>all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very much |
|---|---|---|---|---|---|---|
| HI7 | I feel fatigued | 0 | 1 | 2 | 3 | 4 |
| HI12 | I feel weak all over | 0 | 1 | 2 | 3 | 4 |
| An1 | I feel listless ("washed out") | 0 | 1 | 2 | 3 | 4 |
| An2 | I feel tired | 0 | 1 | 2 | 3 | 4 |
| An3 | I have trouble starting things because I am tired | 0 | 1 | 2 | 3 | 4 |
| An4 | I have trouble <u>finishing</u> things because I am tired | 0 | 1 | 2 | 3 | 4 |
| An5 | I have energy | 0 | 1 | 2 | 3 | 4 |
| An7 | I am able to do my usual activities | 0 | 1 | 2 | 3 | 4 |
| An8 | I need to sleep during the day | 0 | 1 | 2 | 3 | 4 |
| An12 | I am too tired to eat | 0 | 1 | 2 | 3 | 4 |
| An14 | I need help doing my usual activities | 0 | 1 | 2 | 3 | 4 |
| An15 | I am frustrated by being too tired to do the things I want to do | 0 | 1 | 2 | 3 | 4 |
| An16 | I have to limit my social activity because I am tired | 0 | 1 | 2 | 3 | 4 |

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL - 

## **FACIT-Fatigue Subscale Scoring Guidelines** (Version 4)

- Instructions:\* 1. Record answers in "item response" column. If missing, mark with an X
  - 2. Perform reversals as indicated, and sum individual items to obtain a score.
  - 3. Multiply the sum of the item scores by the number of items in the subscale, then divide by the number of items answered. This produces the subscale score.
  - 4. The higher the score, the better the QOL.

| <b>Subscale</b> | Item Code | Revers | se item? | <u>Item response</u> | <b>Item Score</b> |
|---|---|---|---|---|---|
| FATIGUE | HI7 | 4 | _ | | = |
| <b>SUBSCALE</b> | HI12 | 4 | - | | = |
| | An1 | 4 | - | | = |
| | An2 | 4 | - | | = |
| Score range: 0-52 | An3 | 4 | - | | = |
| 2000 m.gev v v= | An4 | 4 | - | | = |
| | An5 | 0 | + | | = |
| | An7 | 0 | + | | = |
| | An8 | 4 | - | | = |
| | An12 | 4 | - | | = |
| | An14 | 4 | - | | = |
| | An15 | 4 | - | | = |
| | An16 | 4 | - | | = |
| Sum individual | item scores: | | | _ | |
| Multiply by 13: | | | | | |
| Divide by num | ber of items | | | | |
| answered: | | | | _ (Fatigue Subscale | Score) |

<sup>\*</sup>For guidelines on handling missing data and scoring options, please refer to the Administration and Scoring Guidelines in the manual or on-line at www.facit.org.

NOTE: The FACIT and all related works are owned and copyrighted by, and the intellectual property of David Cella, Ph.D. Permission for use of the FACIT-FATIGUE questionnaire is obtained by contacting Dr. Cella at information@facit.org

Apellis Pharmaceuticals, Inc. - CONFIDENTIAL -

#### 16. APPENDIX 2: LASA SCALE

## LINEAR ANALOG SCALE ASSESSMENT

Three questions about how you felt during this past week are listed below. Please place a **VERTICAL** mark on the line to indicate your answer. The position of the mark, somewhere between the two extremes, should reflect how you feel.







